# STATISTICAL ANALYSIS PLAN

# A PHASE 2 TRIAL OF NIROGACESTAT IN PATIENTS WITH RECURRENT OVARIAN GRANULOSA CELL TUMORS

Protocol Number: NIR-OGT-201

**Protocol Version and Date:** Amendment 5: 19Mar2024

Amendment 4: 07Jun2023 Amendment 3: 31Jan2023 Amendment 2: 18Jul2022 Amendment 1: 12Dec2021

Original: 09Nov2021

Name of Test Drug: Nirogacestat

Phase: Phase II

**Sponsor:** SpringWorks Therapeutics

100 Washington Blvd.

Stamford, CT 06902

United States

**Authors:** Carmelita Alvero/Steven Chang

Analysis Plan Date: 28Oct2024

Analysis Plan Version: Version 3.0

### **Confidentiality Statement**

The information in this document is confidential information of SpringWorks Therapeutics and is not to be disclosed without the prior written consent of SpringWorks. You are allowed to disclose the contents of this document only to study personnel directly involved with conducting this study and who are bound by obligations of confidentiality in connection with their involvement with this study. Persons to whom the information is disclosed must be informed that the information is confidential and proprietary to SpringWorks and that it may not be further disclosed to third parties or used for any other purpose. The disclosure and use of information in this document are subject to a written confidentiality agreement between SpringWorks and your organization.



# **APPROVALS**

| Signed by: | |
|---|---|
| Steven Chang | |
| Signer Name: Steven Chang Signing Reason: I am the author of this document | |
| Signing Time: 29-Oct-2024 10:41:56 EDT | 29-Oct-2024 10:42:29 EDT |
| 32411558E40F490F83BD132F2BF65799 | 29-0Ct-2024 10.42.29 EDT |
| Steven Chang | Date |
| Statistical Consultant, Biostatistics | |
| SpringWorks Therapeutics, Inc. | |
| Signed by: | |
| Carmelita Alvero | |
| Circus Names Cormolite Alvers | |
| Signer Name: Carmelita Alvero Signing Reason: I am the author of this document | |
| Signing Time: 29-Oct-2024 10:38:01 EDT | 29-Oct-2024 10:38:22 EDT |
| FC9A702759074B62B0EB8FAC79DE2641 | 20 100 2121 20101122 221 |
| Carmelita Alvero | Date |
| Associate Director, Biostatistics | |
| SpringWorks Therapeutics, Inc. | |
| Approver Signatories: | |
| Approver Signatories: | |
| Signed by: | |
| Signed by: Joulyn Liwis Signer Name: Jocelyn Lewis | |
| Signed by: Joulyn Lewis | |
| Signed by: Signer Name: Jocelyn Lewis Signing Reason: I approve this document | 31-Oct-2024 09:59:28 EDT |
| Signed by: Joulyn Lwis Signer Name: Jocelyn Lewis Signing Reason: I approve this document Signing Time: 31-Oct-2024 09:58:59 EDT D920FBC6135E4F3A9DE7358EDE3C6954 | |
| Signed by: Jouly Liwis Signer Name: Jocelyn Lewis Signing Reason: I approve this document Signing Time: 31-Oct-2024 09:58:59 EDT D920FBC6135E4F3A9DE7358EDE3C6954 Jocelyn Lewis | 31-oct-2024 09:59:28 EDT Date |
| Signed by: Jouly Livis Signer Name: Jocelyn Lewis Signing Reason: I approve this document Signing Time: 31-Oct-2024 09:58:59 EDT D920FBC6135E4F3A9DE7358EDE3C6954 Jocelyn Lewis Medical Director, Clinical Development | |
| Signed by: July Lwis Signer Name: Jocelyn Lewis Signing Reason: I approve this document Signing Time: 31-Oct-2024 09:58:59 EDT D920FBC6135E4F3A9DE7358EDE3C6954 Jocelyn Lewis Medical Director, Clinical Development SpringWorks Therapeutics, Inc. | |
| Signed by: July Liwis Signer Name: Jocelyn Lewis Signing Reason: I approve this document Signing Time: 31-Oct-2024 09:58:59 EDT D920FBC6135E4F3A9DE7358EDE3C6954 Jocelyn Lewis Medical Director, Clinical Development SpringWorks Therapeutics, Inc. Signed by: | |
| Signed by: July Lwis Signer Name: Jocelyn Lewis Signing Reason: I approve this document Signing Time: 31-Oct-2024 09:58:59 EDT D920FBC6135E4F3A9DE7358EDE3C6954 Jocelyn Lewis Medical Director, Clinical Development SpringWorks Therapeutics, Inc. | |
| Signed by: July Lwis Signer Name: Jocelyn Lewis Signing Reason: I approve this document Signing Time: 31-Oct-2024 09:58:59 EDT D920FBC6135E4F3A9DE7358EDE3C6954 Jocelyn Lewis Medical Director, Clinical Development SpringWorks Therapeutics, Inc. Signed by: Signer Name: Steven Hege | |
| Signed by: July Lwis Signer Name: Jocelyn Lewis Signing Reason: I approve this document Signing Time: 31-Oct-2024 09:58:59 EDT D920FBC6135E4F3A9DE7358EDE3C6954 Jocelyn Lewis Medical Director, Clinical Development SpringWorks Therapeutics, Inc. Signed by: Sturn Han | |
| Signed by: July Lwis Signer Name: Jocelyn Lewis Signing Reason: I approve this document Signing Time: 31-Oct-2024 09:58:59 EDT D920FBC6135E4F3A9DE7358EDE3C6954 Jocelyn Lewis Medical Director, Clinical Development SpringWorks Therapeutics, Inc. Signed by: Junt Han Signer Name: Steven Hege Signing Reason: I approve this document | Date |
| Signed by: July Liwis Signer Name: Jocelyn Lewis Signing Reason: I approve this document Signing Time: 31-Oct-2024 09:58:59 EDT D920FBC6135E4F3A9DE7358EDE3C6954 Jocelyn Lewis Medical Director, Clinical Development SpringWorks Therapeutics, Inc. Signed by: Signer Name: Steven Hege Signing Reason: I approve this document Signing Time: 31-Oct-2024 11:42:14 EDT | |
| Signed by: July Lwis Signer Name: Jocelyn Lewis Signing Reason: I approve this document Signing Time: 31-Oct-2024 09:58:59 EDT D920FBC6135E4F3A9DE7358EDE3C6954 Jocelyn Lewis Medical Director, Clinical Development SpringWorks Therapeutics, Inc. Signed by: Signer Name: Steven Hege Signing Reason: I approve this document Signing Time: 31-Oct-2024 11:42:14 EDT C575696753774E0DAFD1AB6D72356E5C | Date |
| Signed by: July Liwis Signer Name: Jocelyn Lewis Signing Reason: I approve this document Signing Time: 31-Oct-2024 09:58:59 EDT D920FBC6135E4F3A9DE7358EDE3C6954 Jocelyn Lewis Medical Director, Clinical Development SpringWorks Therapeutics, Inc. Signed by: Signer Name: Steven Hege Signing Reason: I approve this document Signing Time: 31-Oct-2024 11:42:14 EDT | Date 31-oct-2024 11:42:40 EDT |



# Contents

| 1. | SUMMARY OF STUDY PROTOCOL | 9 |
|---|---|---|
| 1.1. | Introduction and Study Rationale | 9 |
| 1.2. | Study Objectives and Endpoints | 10 |
| 1.3. | Study Design | 12 |
| 1.4. | Sample Size Determination | 13 |
| 1.5. | Data Monitoring Committee | 16 |
| 2. | Analysis Sets | |
| 2.1. | Analysis Set Definitions | 17 |
| 2.2. | Protocol Deviations | 17 |
| 2.3. | Impacts from COVID-19 | 17 |
| 3. | ENDPOINTS | 19 |
| 3.1. | Primary Efficacy Endpoint | 19 |
| 3.2. | Secondary Efficacy Endpoints | 19 |
| 3.3. | Exploratory Efficacy Endpoints | 19 |
| | Safety Endpoints | |
| 3.5. | Pharmacokinetic Endpoints | 20 |
| 3.6. | Other Endpoints | 20 |
| 4. | STATISTICAL METHODOLOGY | 21 |
| 4.1. | General Information | 21 |
| 4.2. | Baseline Definitions | 22 |
| 4.3. | Methods of Pooling Data | 22 |
| 4.4. | Adjustments for Covariates | 22 |
| 4.5. | Multiple Comparisons/Multiplicity | 22 |
| | Subgroups | |
| 4.7. | Withdrawals, Dropouts, Loss to Follow-up. | 23 |
| 4.8. | Missing Data Conventions for Efficacy Endpoints | 23 |
| 4.9. | Missing Data Conventions for Safety Endpoints | 23 |
| 4.9.1 | Handling of Missing/Partial Dates for AEs | 23 |
| 4.9.2 | 2. Handling of Concomitant Therapies/Medications with Missing/Partial Dates | 24 |
| 4.9.3 | 3. Handling of Missing Dates for Disease History and Prior Therapies | 24 |
| 4.10 | . Visit Windows | |
| 5. | STATISTICAL ANALYSES | 26 |
| | Disposition | |
| 5.2. | Demographics, Baseline Characteristics, and Medical History | 27 |
| 5.2.1 | Demographics | 27 |
| 5.2.2 | <b>→</b> | |
| 5.2.3 | 3. Medical History | 27 |
| 5.2.4 | | |
| 5.3. | Primary Efficacy Endpoint. | |
| 5.3.1 | , | |
| 5.3.2 | , | |
| 5.3.3 | | |
| | Secondary Efficacy Endpoints | |
| 5.4.1 | | |
| 5.4.2 | 2. OS-2 | 29 |



| 5.4.3. | Change from Baseline in FOSI-8 | 30 |
|---|---|---|
| 5.4.4. | Duration of Response (DoR) | 30 |
| 5.5. Explo | pratory Efficacy Endpoints | 31 |
| 5.5.1. | Time to Event Endpoints | 31 |
| 5.5.2. | Next Generation Sequencing status | 33 |
| 5.5.3. | Inhibin A&B, Follicle-stimulating Hormone, Estradiol, CA-125, and AMH/Mullerian Inhib | |
| Substance | (MIS) | 33 |
| 5.5.4. | Time to Response | |
| 5.6. Safety | Analyses | |
| 5.6.1. | Study Dug Exposure and Compliance | |
| 5.6.2. | Adverse Events | |
| 5.6.3. | Safety Topics of Special Interest | |
| 5.6.4. | Protocol-Required Laboratory Assessments. | |
| 5.6.5. | Physical Exam and Eastern Cooperative Oncology Group Performance Status | |
| 5.6.6. | Electrocardiogram | |
| 5.6.7. | Vital Signs | 42 |
| 5.6.8. | Concomitant Medications | 43 |
| 5.7. Pharm | nacokinetic and Pharmacodynamic Analyses | 44 |
| 5.8. Interi | m Analysis | 44 |
| 6. Chan | NGES TO PLANNED ANALYSES | 48 |
| 7. Refe | RENCES | 49 |
| 8. Appe | NDICES | 51 |
| | ST Criteria V1.1 | |
| 8.2. FACT | T/NCCN Ovarian Symptom Index (FOSI) - Version 4 | 55 |
| 8.3. Mock | -up Tables, Listings, and Figure | 56 |
| 8.4. Safety | Topics of Special Interest Preferred Terms | 56 |
| 8.4.1. | Protocol-Specified AESIs | 56 |
| 8.4.1.1. | Hypersensitivity | 56 |
| 8.4.1.2. | Skin Disorder and Rash | 58 |
| 8.4.1.3. | Hepatotoxicitiy | 60 |
| 8.4.1.4. | Electrolyte Disorder | 66 |
| 8.4.1.5. | Non-Melanoma Skin Cancers | 67 |
| 8.4.2. | Other Safety Topics of Special Interest | 68 |
| 8.4.2.1. | Musculoskeletal Disorders | 68 |
| 8.4.2.2. | Bone Fracture | 69 |
| 8.4.2.3. | Mucositis/Stomatitis | 71 |
| 8.4.2.4. | Hematologic Disorders | 71 |
| 8.4.2.5. | Opportunistic Infections | 73 |
| 8.4.2.6. | Central Nervous System Vascular Disorders | 93 |
| 8.4.2.7. | Embolic and Thrombotic Events | |
| 8.4.2.8. | Cardiac Rhythm Disturbances | 98 |
| 8.4.2.9. | Upper Respiratory Tract Infections | |
| 8.4.2.10. | Diarrhea | 99 |
| Plan Versi | on History | |
| | istory Summary | 100 |



# LIST OF TABLES

| Table 1 | Simulated Probability of Early Stopping under Assumed ORR |
|---------|--------------------------------------------------------------|
| Table 2 | Exact 95% CI Given Observed ORR |
| Table 3 | PFS and DoR Censoring Rules |
| Table 4 | Eastern Cooperative Oncology Group Performance Status Grades |



### LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|--------------|------------------------------------------------|
| ADL | Activities of Daily Living |
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ALT | Alanine Aminotransferase |
| AMH | Anti-Mullerian Hormone |
| AST | Aspartate Aminotransferase |
| ATC | Anatomic Therapeutic Class |
| BID | Twice daily |
| BMI | Body Mass Index |
| C | Cycle |
| CA 125 | Cancer Antigen 125 |
| CI | Confidence Interval |
| $C_{max}$ | Maximum plasma concentration |
| $C_{trough}$ | Plasma trough concentration |
| COVID-19 | Coronavirus Disease 2019 |
| CR | Complete response |
| CRF | Case report form |
| CSR | Clinical Study Report |
| CT | Computed tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| ctDNA | Circulating tumor DNA |
| D | Day |
| DNA | Deoxyribonucleic acid |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic case report form |
| EOT | End of Treatment |
| FDA | Food and Drug Administration |



FOSI Functional Assessment of Cancer Therapy – Ovarian Symptom

Index

FSH Follicle-stimulating hormone

FUP Follow-up

GCT Granulosa cell tumors

GOG Gynecologic Oncology Group

HBV Hepatitis B virus

HLGT High Level Group Term

HR Heart rate

ICF Informed Consent Form

INR International normalized ratio

K-M Kaplan-Meier

LD Longest diameter

LH Luteinizing Hormone

MIS Mullerian Inhibiting Substance
MRI Magnetic Resonance Imaging

NE Not evaluable

NGS Next Generation Sequencing

NICD Notch Intracellular Domain

No. Number

ORR Objective Response Rate

OS Overall survival

OS-2 Overall survival probability at 2 years

OvGCTs Ovarian granulosa cell tumors

PD Progressive Disease or Pharmacodynamics

PFS Progression free survival

PFS2 Progression free survival 2

PFS-6 Progression-free survival at 6 months

PK Pharmacokinetics

PR Partial Response

QRS QRS complex



QT Uncorrected QT interval

QTc Corrected QT interval

QTcF Corrected QT interval by Fredericia

RECIST Response Evaluation Criteria in Solid Tumors

SAE Serious adverse event

SAP Statistical Analysis Plan

SD Stable disease

SoA Schedule of Assessments

SOC System Organ Class

TEAE Treatment Emergent Adverse Event

ULN Upper Limit of Normal



### 1. SUMMARY OF STUDY PROTOCOL

# 1.1. Introduction and Study Rationale

This document is the statistical analysis plan (SAP) for NIR-OGT-201, a Phase 2 trial of nirogacestat in Patients with Recurrent Ovarian Granulosa Cell Tumors study to assess the antitumor activity of nirogacestat in adult participants with relapsed/refractory ovarian granulosa cell tumors (OvGCTs). Standard of care treatment for relapsed/refractory OvGCT is platinum-based chemotherapy consisting of bleomycin, etoposide, and cisplatin or carboplatin and paclitaxel. These chemotherapy regimens, however, are not associated with durable remissions and most participants eventually develop progressive disease necessitating treatment with experimental agents. In prior studies in progressive OvGCTs, experimental agents have shown promise with only modest performance. In the Gynecologic Oncology Group (GOG) study of bevacizumab monotherapy, the Objective Response Rate (ORR) was 16.7% with a median Progression Free Survival (PFS) of 9.3 months (Brown et al. 2014). Combination therapy of bevacizumab with paclitaxel showed an improved ORR of 44% compared to 25% for paclitaxel monotherapy but did not improve PFS (Ray-Coquard et al. 2020).

Our hypothesis is that treatment of relapsed/refractory OvGCT with nirogacestat 150 mg twice daily (BID) will provide at least ORR of 30% with a secondary objective of improved duration of PFS and Overall Survival (OS) compared to bevacizumab monotherapy. In order to limit accrual of participants to ineffective treatments, the study will use a Bayesian strategy (J. Lee and Liu 2008; Chen et al. 2019) for continuous futility monitoring for early stopping based on ORR. Bayesian predictive probability will be used throughout the trial to assess the posterior probability of obtaining an ORR of no less than 15%.

Treatment of granulosa cell tumors with a gamma secretase (GS) inhibitor such as nirogacestat is expected to inhibit Notch-induced granulosa cell proliferation by (1) limiting activation of growth factor signaling by the FOXL2 mutant protein, (2) inhibiting proliferation signaling through NICD and (3) by inducing apoptosis through the pAKT activation.

This SAP further details the statistical analyses to be conducted during and at the end of the study as determined in the protocol. It is designed to outline the methods to be used in the



analysis of study data to achieve the study objective(s). Populations for analysis, data handling rules, statistical methods, and formats for data presentation are provided. The statistical analyses and summary tabulations described in this SAP will provide the basis for the results sections of the clinical study report (CSR) for this trial.

This SAP will also outline any differences in the currently planned analytical objectives relative to those planned in the study protocol if there is any.

# 1.2. Study Objectives and Endpoints

The study objectives and corresponding analysis endpoints are listed below.

| Primary Objectives: | Primary Endpoints: |
|---|---|
| To determine the anti-tumor activity of nirogacestat in adult participants with relapsed/refractory OvGCT | Objective response rate (ORR), defined as<br>the proportion of participants with Complete<br>Response (CR) + Partial Response (PR)<br>using Response Evaluation Criteria in Solid<br>Tumors (RECIST) v1.1 |
| Secondary Objectives: | Secondary Endpoints: |
| To determine if nirogacestat delays progression or death in OvGCT | Estimate of proportion of participants who have not progressed or died at 6 months follow-up: PFS-6. Progression is defined by RECIST v1.1 |
| To describe overall survival in participants treated with nirogacestat | Estimate of 2-year overall survival, defined as the proportion of participants who have not died after 2 years of follow-up after their first dose of nirogacestat |
| To determine the effect of nirogacestat on ovarian cancer symptoms measured by Functional Assessment of Cancer Therapy – Ovarian Symptom Index (FOSI) | Change from baseline in FOSI |
| To determine the duration of response | Duration of response (DoR), defined as the time from first assessment of response (CR + PR using RECIST v1.1) to first disease progression defined by RECIST v1.1 or death, whichever comes first |



| To determine the pharmacokinetics (PK) of nirogacestat | Serum concentrations of nirogacestat will be measured to evaluate system exposures (Cmax, Ctrough and other PK parameters as data allow) |
|---|---|
| Safety Objectives | Safety Endpoints |
| To characterize the safety and tolerability of nirogacestat at a dose of 150 mg BID in adult participants with relapsed/refractory OvGCT | Key safety endpoints will include incidence of treatment-emergent Adverse Events (TEAEs), changes in clinical laboratory parameters, vital signs, physical examination findings, and electrocardiograms (ECGs) Tolerability will be assessed according to toxicities graded by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0 |
| <b>Exploratory Objectives</b> | Exploratory Endpoints |
| To detect FOXL2 C134W mutation as well as other genomic alterations and correlate these with response | Evaluate Next Generation Sequencing (NGS) status in baseline tumor tissue |
| To detect NICD and candidate biomarkers of response, and to correlate nirogacestat exposure with response | <ul> <li>Evaluate change from Baseline:</li> <li>Inhibin A&amp;B, Follicle-stimulating hormone (FSH), estradiol, CA-125, and Mullerian Inhibiting Substance (MIS) / AMH</li> <li>Circulating tumor DNA (ctDNA)</li> <li>Baseline NICD expression in tumor tissue</li> </ul> |
| To describe progression free survival on continued nirogacestat treatment post first disease progression | Progression free survival on prolonged nirogacestat treatment, defined as time from first disease progression per RECIST v1.1 to second disease progression on continued nirogacestat treatment confirmed by investigator discretion or death, whichever comes first |



| To describe progression free survival on | Progression free survival 2 (PFS2), defined as |
|---|---|
| subsequent line of anticancer treatment | time from first dose of nirogacestat to second |
| | disease progression on subsequent line of |
| | anticancer treatment (after nirogacestat) |
| | confirmed by investigator discretion at long |
| | term safety follow-up visit or death, |

whichever comes first.

### 1.3. Study Design

This is a multi-center, single-arm, Phase 2 open label treatment study to determine the efficacy, safety, tolerability, and pharmacokinetics of nirogacestat in adult participants with recurrent OvGCT. Participants must have received at least one prior course of systemic therapy for OvGCT and have measurable disease by RECIST v1.1 to meet the eligibility criteria.

The Schedule of Assessments (SoA) is in protocol Section 1.3, Table 2. Participants will be screened up to 28 days prior to the first dose of study treatment (nirogacestat) and full eligibility will be based on the inclusion and exclusion criteria (Protocol Section 7.1 and 7.2).

Participants will administer 150 mg ( $3 \times 50 \text{ mg}$  tablets) of study treatment BID, continuously in 28-day cycles. Participants will remain on study treatment until death, disease progression (unless the participants meet criteria for continued treatment), discontinuation of study treatment for any reason, the study is stopped by the Sponsor for any reason, or participant qualifies for Sponsor's Compassionate Use Program.

All scans will be performed and read locally by the site's radiologist for Tumor assessment as per RECIST v1.1. Same modality used at Screening must be used at each subsequent imaging visits. Baseline scan is defined as scans performed prior to first dose of study treatment. On treatment scans are performed every 8 weeks (C3D1, C5D1, C7D1) for the first 6 months and then every 12 weeks (C10D1, C13D1, etc.) thereafter. Scans may be performed (-) 7 days prior to the visit.

The final 2-year survival check-in will occur approximately 2 years after the first dose of study treatment. If participant discontinues from study treatment prior to the 2-year check-in, quarterly telephone or email contact following EOT is required until the 2-year survival data point has



been collected. In addition, collection of subsequent anticancer therapy after nirogacestat and overall response to this therapy will be recorded. Only information about the subsequent therapy used directly after nirogacestat is required along with the final survival outcome at the 2-year check point.

Participants who discontinue study treatment early for any reason should return to the clinic for an End of Treatment (EOT) visit within 7 days after the Investigator determines study treatment will no longer be used and then again for a safety Follow-up (FUP) visit 30 days (+7 days) after the last dose of study treatment.

The estimated study duration is 3 years, and all participants will be followed for at least 2 years (unless the study is prematurely stopped due to futility).

A Bayesian strategy allowing continuous monitoring will be used to evaluate the posterior distribution of ORR (complete + partial) (<u>Lee and Liu 2008</u>; <u>Chen et al. 2019</u>) and the study may be stopped for futility if necessary. There will be no pause in accrual for interim assessments.

# 1.4. Sample Size Determination

A prior GOG phase 2 trial in previously treated participants with stromal tumors evaluated the efficacy and safety of bevacizumab monotherapy in participants with recurrent sex cord stromal tumors of the ovary. The ORR in this study was 16.7% (Brown et al. 2014). Following this outcome, the ALIENOR/ENGOT ov7 trial randomized participants to see if the addition of bevacizumab to paclitaxel had effect on the PFS rate among participants with relapsed ovarian sex cord stromal tumors. While the combination therapy of paclitaxel and bevacizumab showed an ORR of 44% over paclitaxel monotherapy, the PFS remained equivocal between the two treatment groups (Ray-Coquard et al. 2020). Based on the ORR from the bevacizumab monotherapy trial, this study aims for an ORR of 30% with PFS as a secondary endpoint.

Since this is a first-in-human proof of concept study for the indication, no formal hypothesis testing or sample size calculation is contemplated. The initial goal of accrual for this study is 43 participants which should provide sufficient sample size for interim evaluations for futility with a Bayesian strategy of continuous monitoring. Participant accrual will not be paused during the interim evaluations. The Bayesian approach to be used for futility analysis assumes a



beta-binomial distribution with an uninformative prior of beta distribution (Lee and Liu 2008; Chen et al. 2019). Assume at an assessment point, the study has accrued X responders out of n ( $\leq$ 43) participants. With a prior distribution of *beta* (a, b), X follows a binomial distribution and the posterior distribution of the response rate follows a beta distribution with parameters (a+x, b+n-x), where x is the observed value of X. Thus, the number of responses in the potential (43-n) future participants, Y, follows a beta-binomial distribution with parameters (43-n, a+x, b+n-x). From the observed responders x and a target ORR, the predictive probability of reaching the target ORR at the end of study can be calculated with the beta-binomial distribution. If the predictive probability is too low, e.g.,  $\leq$ 10%, the study may be terminated for futility. A high predictive probability, e.g.,  $\geq$ 85%, suggests high likelihood of achieving treatment efficacy at the end of the study.

For this study, we assume that a response rate of  $\leq$ 15% at the end of study is considered ineffective for the treatment, and enrollment will stop if the posterior probability of ORR >15% is less than 0.1. On the other hand, the treatment is considered promising if the posterior probability of ORR >15% is higher than 0.85, that is, if the posterior distribution provides

$$Prob\{ORR > 0.15 | data\} > 0.85.$$

For calculating the posterior probability, a prior of beta (0.1, 0.9) could be assumed. These parameters (0.1 and 0.9) of the beta prior correspond to the initial assumed distribution of ORR with mean equal to 0.1/(0.1+0.9) = 10% (that is, an initial belief of ORR around 10%). The beta parameters will be updated according to observed number of responders at each analysis.

Given the cutoff points of the predictive probability for futility and efficacy, the characteristics of the design can be assessed in terms of type I and II errors. For example, if the cutoff points are set at 10% for futility and 85% for efficacy, the above Bayesian rule will result in futility stopping boundaries of 1, 2, and 5 or fewer respondents if interim evaluations were to occur at enrollment of 10, 20, 30 participants, respectively. If the true rate of ORR is 15%, the chance to conclude treatment efficacy at the end of the study is 7% (Type I error). However, the probability to stop the trial early is 79%. If the true rate of ORR is 30%, the chance to conclude treatment efficacy at the end of the study is 76%.



A set of simulations using a frequentist framework under the similar interim evaluation schedule as above are performed for comparisons. Specifically, the type I and II errors are simulated for scenarios where the study ceases for futility when the ORRs are 0%,  $\leq 5\%$ ,  $\leq 10\%$ , or 15% when 10, 20, 30, and 43 participants have been enrolled, respectively. Those conditions correspond to stopping for futility when there are fewer than or equal to 0, 1, 3, and 6 respondents in the three interim and final analyses, respectively. Table 1 below provides results based on 10,000 simulations of probability of early stopping for futility and the expected overall sample sizes.

Table 1 Simulated Probability of Early Stopping under Assumed ORR

| Interim Tin<br>(Enrollmen | | 10 | 20 | 30 | 43 | | | Efficacy | Average |
|---|---|---|---|---|---|---|---|---|---|
| Stopping Bo<br>(No. of Resp | | | 1 | 3 | Futility at First Three 6 Looks | | Futility at<br>End of<br>Study | at End of Study | Overall<br>Sample<br>Size <sup>1</sup> |
| ., <b>~</b> | 0.05 | 0.60 | 0.19 | 0.16 | 0.05 | 0.95 | 1.00 | 0.00 | 11 |
| True<br>3 ORR | 0.10 | 0.35 | 0.13 | 0.21 | 0.19 | 0.69 | 0.88 | 0.12 | 22 |
| | 0.15 | 0.20 | 0.07 | 0.13 | 0.19 | 0.40 | 0.59 | 0.41 | 32 |
| ume<br>rlyj | 0.20 | 0.11 | 0.03 | 0.06 | 0.10 | 0.20 | 0.30 | 0.70 | 38 |
| Assumed T | 0.25 | 0.06 | 0.01 | 0.02 | 0.03 | 0.09 | 0.12 | 0.88 | 41 |
| , D | 0.30 | 0.03 | 0.00 | 0.01 | 0.01 | 0.04 | 0.04 | 0.96 | 42 |

ORR = Objective Response Rate, N = Sample size; No. = Number

As can be seen from the above table, the probabilities to stop for futility early if true ORR is either 5% or 10% are approximately 100% and 88%, respectively. The probabilities to stop for futility when true ORR is either 25% or 30% are approximately 12% and 4%, respectively. For various criteria to claim efficacy, the exact 95% CI for different corresponding observed ORR based on the Clopper-Pearson method are listed in Table 2. For example, if the total sample size is 20 at the second interim evaluation, the lower bound of the 95% CI will be 27.2% if the observed ORR is 50%. When the total sample size is 30 or higher and the observed ORR is 50%, the lower bound of the 95% CI will be  $\geq$ 31.3%.

<sup>&</sup>lt;sup>1</sup>Without considering newly enrolled participants while the interim evaluation is ongoing.



Table 2 Exact 95% CI Given Observed ORR

| Minimum ORR | Observed No. | Observed ORR | 95% Confidence Interval | | |
|---|---|---|---|---|---|
| to Claim Efficacy | Sample Size | of Responders | (%) | Lower<br>Bound | Upper<br>Bound |
| 0.25 | 10 | 3 | 30.0 | 6.7 | 65.3 |
| | 20 | 5 | 25.0 | 8.7 | 49.1 |
| | 30 | 8 | 26.7 | 12.3 | 45.9 |
| | 43 | 11 | 25.6 | 13.5 | 41.2 |
| 0.3 | 10 | 3 | 30.0 | 6.7 | 65.3 |
| | 20 | 6 | 30.0 | 11.9 | 54.3 |
| | 30 | 9 | 30.0 | 14.7 | 49.4 |
| | 43 | 13 | 30.2 | 17.2 | 46.1 |
| 0.5 | 10 | 5 | 50.0 | 18.7 | 81.3 |
| | 20 | 10 | 50.0 | 27.2 | 72.8 |
| | 30 | 15 | 50.0 | 31.3 | 68.7 |
| | 43 | 22 | 51.2 | 35.5 | 66.7 |

CI = Confidence Interval; ORR = Objective Response Rate

# 1.5. Data Monitoring Committee

There is no Data Monitoring Committee for this study.



### 2. ANALYSIS SETS

# 2.1. Analysis Set Definitions

The following participant analysis sets will be evaluated and used for presentation and analysis of the data:

- Screened Analysis Set: The Screened Analysis Set will consist of all participants who signed the informed consent.
- Full Analysis Set: The Full Analysis Set will consist of all participants who received at least 1 dose of nirogacestat treatment.
- PK Analysis Set: The PK Analysis Set will consist of all treated participants with at least 1 non-missing value in serum concentration of nirogacestat.
- Safety Analysis Set: The Safety Analysis Set will consist of all participants who received at least 1 dose of nirogacestat treatment.

The Full Analysis Set is the same as the Safety Analysis Set. All efficacy analyses will be based on the Full Analysis Set. All safety analyses will be based on the Safety Analysis Set.

### 2.2. Protocol Deviations

Protocol deviations are reviewed in accordance with the Protocol Deviation Management Plan. All Major and Minor protocol deviations will be reviewed by SpringWorks prior to database lock. The protocol deviation categories are defined in the Protocol Deviation Management Plan, including those related to the inclusion/exclusion criteria, informed consent, withdrawal criteria, study treatment, etc. Major protocol deviations and the COVID-19 related major protocol deviations will be summarized. A data listing of all PDs including a description of the deviation will be generated, and the COVID-19 related protocol deviations will be flagged.

# 2.3. Impacts from COVID-19

This study was conducted during the global SARS-Cov-2 pandemic. The impact of COVID-19 was mitigated based on the evolving EMA and FDA COVID-19 guidelines [European Medicines Agency 2021; US Food and Drug Administration 2020].



A listing of all participants impacted by COVID-19 and how their participation in the study was altered, including missed visits, missed assessments, impacts on the tumor assessments, and other deviations from protocol procedures due to COVID-19 will be provided.



### 3. ENDPOINTS

# 3.1. Primary Efficacy Endpoint

The primary efficacy endpoint is objective response rate, defined as the proportion of participants with CR + PR using RECIST v1.1. See Section 8.1 for the details of RECIST Criteria v1.1.

Study participants who have no post-baseline tumor assessment and those whose best overall response is not evaluable or less than CR or PR will be analyzed as a non-responder.

# 3.2. Secondary Efficacy Endpoints

Secondary efficacy endpoints include:

- PFS-6, defined as the survival probability of not having progressed or died at 6 months follow-up. Progression is defined by RECIST v1.1.
- Two-year overall survival at 2 years (OS-2), defined as the survival probability of being still alive at 2 years of follow-up after their first dose of nirogacestat.
- Change from baseline in FOSI.
- DoR, defined as the time from first assessment of response (CR + PR using RECIST v1.1) to first disease progression defined by RECIST v1.1 or death, whichever comes first.

# 3.3. Exploratory Efficacy Endpoints

Exploratory endpoints include:

- Progression free survival (PFS), defined as time from first dose of nirogacestat to first disease progression on nirogacestat or death from any cause, whichever comes first.
- Progression free survival on continued nirogacestat treatment, defined as time from first
  disease progression per RECIST v1.1 to second disease progression on continued
  nirogacestat treatment confirmed by investigator discretion or death, whichever comes
  first.
- Progression free survival 2 (PFS2), defined as time from first dose of nirogacestat to second disease progression on subsequent line of anticancer treatment (after nirogacestat)



confirmed by investigator discretion at long term safety follow-up visit or death, whichever comes first.

- Overall survival (OS), defined as time from first dose of nirogacestat to death from any cause.
- Time to response, defined as time in months from first dose until date of the first documented response (CR or PR).
- Evaluate Next Generation Sequencing (NGS) status in baseline tumor tissue.
- Change from baseline in:
  - Inhibin A&B, Follicle-stimulating, hormone (FSH), estradiol, CA-125, and Mullerian
     Inhibiting Substance (MIS) / AMH
  - o Circulating tumor DNA (ctDNA) (if data are available)
- Baseline NICD expression in tumor tissue (if data are available).

# 3.4. Safety Endpoints

Key safety endpoints will include incidence of treatment-emergent Adverse Events (TEAEs), changes in clinical laboratory parameters, vital signs, physical examination findings, and electrocardiograms (ECGs).

Tolerability will be assessed according to toxicities graded by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

# 3.5. Pharmacokinetic Endpoints

Pharmacokinetic endpoints include C<sub>trough</sub> and 1-hour post-dose serum concentrations of nirogacestat.

# 3.6. Other Endpoints

Not applicable.



### 4. STATISTICAL METHODOLOGY

### 4.1. General Information

All data listings that contain an evaluation date will have a relative study day associated with treatment start (Rel Day). Pre-treatment and on-treatment study days represented as Relative Day are numbered relative to the day of the first dose of study medication which is designated as Day 1. The preceding day is Day -1, the day before that is Day -2, etc.

Tabulations will be produced for appropriate disposition, demographic, baseline characteristics, efficacy, and safety parameters. For categorical variables, summary tabulations of the number and percentage of participants within each category (with a category for missing data) of the parameter will be presented. For continuous variables, the number of participants, mean, median, standard deviation, minimum, and maximum values will be presented. Time-to-event data will be summarized using 25<sup>th</sup>, 50<sup>th</sup> (median) and 75<sup>th</sup> percentiles and time point survival probabilities (at 6 months, 1 year, 18 months, 2 years, etc.) with associated 2-sided 95% confidence intervals (CIs) using Kaplan-Meier methodology and the log-log transformation, as well as number and percentage of events and censored observations.

Graphical displays will be provided where useful to aid in the interpretation of results. A swimmer plot may be used to present the exposure to study treatment, overall response and follow up for all participants in the Full Analysis Set. Each participant will be presented on a horizontal bar (y-axis) over time (x-axis) starting at treatment start date. For each participant's bar, the plot will include best overall response (CR, PR, SD, PD, or NE), end of response or continued response (at censored timepoint).

The following conversion conventions will be applied:

- CIs will be presented to 1 more decimal place than the raw data
- Weeks will be calculated as number of days divided by 7
- Months will be calculated as number of days divided by 30.4375
- Years will be calculated as number of days divided by 365.25
- Cycles as used in adverse event summaries are defined as every 28 days
- Day 1 will be considered as the first day of treatment



All tables, figures, and listings will include footers at the bottom of the page reflecting the path of the programs used to generate the tables, figures, and listings, and date and time of the generation of the output.

All descriptive statistical analyses will be performed using SAS statistical software Version 9.4 or higher. Medical history and adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 27.0. Concomitant medications will be coded using the World Health Organization (WHO) Drug Dictionary Version March 2022 or later.

### 4.2. Baseline Definitions

For all analyses, baseline will be defined as the last non-missing value prior to the first administration of study treatment.

# 4.3. Methods of Pooling Data

Data will be pooled across study sites.

# 4.4. Adjustments for Covariates

In this single arm study, covariate adjustment will not be used unless specified otherwise.

# 4.5. Multiple Comparisons/Multiplicity

Since this is a first-in-human proof of concept study for the indication, no formal hypothesis testing is contemplated. Hence there is no multiplicity adjustment for the primary or secondary efficacy endpoints.

# 4.6. Subgroups

Subgroup analyses for the primary endpoint ORR are not predefined due to the following reasons:

- This is a single arm study with a small sample size.
- The anticipated response rate is low-to-medium.

However, post-hoc analysis for subgroup analyses will be performed if deemed necessary.



# 4.7. Withdrawals, Dropouts, Loss to Follow-up

Participants who are withdrawn or discontinue from the study will not be replaced.

# 4.8. Missing Data Conventions for Efficacy Endpoints

There will be no imputation or substitutions made to accommodate missing efficacy data points. All data recorded on the eCRF will be included in data listings that will accompany the CSR.

# 4.9. Missing Data Conventions for Safety Endpoints

# 4.9.1. Handling of Missing/Partial Dates for AEs

Adverse events with incomplete onset dates will be handled as follows for the purpose of determining treatment emergence.

- 1. If the month and day are missing:
  - If the year of the event is the **same** as the year of the first dosing date, then the day and month of the first dosing date will be assigned to the missing fields.
  - If the year is **prior to** the year of first dosing date, then December 31 will be assigned to the missing fields.
  - If the year is **after** the year of first dosing, then January 1 will be assigned to the missing fields.
- 2. If the day is missing:
  - If the month and year are the same as the month of treatment, the onset date will be assigned to the date of treatment.
  - If the month and year are not the same as the month/year of treatment, then the onset day will be set to the first day of the month.

If the start date is completely missing and end date is not before the first dose of study treatment, then the adverse event will be considered treatment emergent.

If the participant has died and the imputed date is later than the date of death, the date of death will be used.



# 4.9.2. Handling of Concomitant Therapies/Medications with Missing/Partial Dates

Concomitant medications are defined in Section 5.6.8. Concomitant therapies/medications with start dates that are completely or partially missing will be handled as follows for the propose of determining concomitance.

- 1. If the start date has the month and year but the day is missing, the therapy will be considered concomitant if the month and year are:
  - a. On or after the month and year of the date of the first dose of study treatment
  - b. On or before the month and year of the date of the last dose of study treatment plus
     30 days
- 2. If the start date has the year, but the day and month are missing, the therapy will be considered concomitant if the year is:
  - a. On or after the year of the date of the first dose of study treatment
  - b. On or before the year of the date of the last dose of study treatment plus 30 days.
- 3. If the start date of concomitant therapies is completely missing and the stop date of concomitant therapies is prior to the date of informed consent, then this therapy will not be considered concomitant.
- 4. If the start date of concomitant therapies is completely or partially missing and the stop date of concomitant therapies is on or after the date of the first dose of study treatment, then the therapy will be considered concomitant.
- 5. If the start date and stop date of concomitant therapies are completely missing, then the therapy will be considered concomitant if the therapy was reported as a concomitant therapy.

# **4.9.3.** Handling of Missing Dates for Disease History and Prior Therapies To calculate time from diagnosis or most recent prior therapy to informed consent, partial/missing dates for diagnosis and last prior therapy completion will be imputed as follows:

• If both day and month are missing and the year is prior to the year of screening, the imputed day and month will be July 1.



- If both day and month are missing and the year is the same as the year of screening, the imputed date will be the middle point between January 1 of the year and the screening date. If the middle point falls between two dates, the first of the two dates will be used.
- If day is missing and the month and year are prior to the month and year of screening, the imputed date will be 15th day of the month.
- If day is missing and the month and year are the same as the month and year of screening, the imputed date will be the middle point between the first date of the month and the screening date. If the middle point falls between two dates, the first of the two dates will be used.
- No imputation will be performed if the year is missing.

### 4.10. Visit Windows

No visit windowing was performed. All visits will be tabulated per the evaluation visit as recorded on the eCRF. Repeat, retest, and unscheduled assessments will not be considered for the calculation of summary statistics and figures, unless assessment qualifies as baseline, or otherwise indicated. These types of assessments will be included in the listings.



### 5. STATISTICAL ANALYSES

# 5.1. Disposition

The total number of participants who were screened (who have signed the informed consent), reasons for screen failure and the number in each study population will be summarized based on the Screened Analysis Set.

The end of treatment status (ongoing/discontinued) together with the primary reason for discontinuing the treatment will be summarized as follows:

- Death
- Disease Progression
- Removal From Study (Investigator/Sponsor Decision)
  - o Adverse Event
  - o Excluded Concomitant Medication or Procedure
  - Compliance (Study Treatment/Study Assessments)
  - New Information/Findings
  - Study/Site is Cancelled
  - Relocation
  - Lost to Follow-Up
  - o Other
- Withdrawal of Consent
- Study Completion
- Other

In addition, the end of study status will be summarized including if a participant is participating in the long-term follow-up.

All treatment and study discontinuation data will be listed. A by-participant data listing of inclusion and exclusion criteria not met will be presented.



# 5.2. Demographics, Baseline Characteristics, and Medical History

Demographics and baseline characteristics will be summarized for the Full Analysis Set. In addition, medical history (including any history of infertility), disease characteristics, prior systemic treatment, radiation and surgery will also be summarized for the Full Analysis Set. Demographic and baseline data, disease characteristics, and prior systemic treatment for each participant will be provided in data listings. In addition, data listings containing the details for prior surgery coded with MedDRA (version 27.0) and prior radiation will be provided.

# 5.2.1. Demographics

Demographics will include univariate statistics for age at time of informed consent (years), baseline weight, baseline height, baseline body mass index (BMI) (kg/m²), baseline FOSI, and categorical summaries for age groups, women of childbearing potential (yes / no), baseline ECOG, race, and ethnicity.

### 5.2.2. OvGCT History and baseline Characteristics

Baseline disease characteristics to be summarized including time (in months) since date of original OvGCT diagnosis to first study treatment, age at the original disease diagnosis, refractory disease (yes/no), time from refractory (months), relapse (yes/no), time from the original relapsed OvGCT diagnosis and the most recent relapse to first study treatment (months), history of prior surgery for OvGCT (yes/no), time (months) since the most recent surgery to first study treatment, prior radiation (yes/no), time (months) since the most recent radiotherapy to first study treatment, prior systemic treatment (yes/no), time (months) since the most recent prior treatment (surgery, radiotherapy and systemic treatment) to first study treatment, number of target lesions, number of non-target lesions, and baseline tumor size, defined as the sum of the target lesion diameters per RECIST v1.1.

# 5.2.3. Medical History

The following medical history will be summarized:

• time in months since last menstrual cycle to first study treatment,



- number and percentage of participants with any history of amenorrhea, menstrual irregularities, or infertility, and
- any clinically significant past or ongoing medical conditions, by MedDRA (version 27.0) System Organ Class (SOC) and Preferred Term (PT).

# 5.2.4. Prior Systemic Therapies for OvGCT

Prior systemic therapies for OvGCT will be coded with WHO Drug March 2022 version or higher and will be summarized by anatomic therapeutic class (ATC) and PT.

Details about each line of treatment, including agents start and stop date, reason for discontinuation, best overall response will be listed. The number of lines of systemic treatment, prior use of Bevacizumab (yes/no), time (months) since most recent Bevacizumab use and time (months) since most recent systemic treatment line to first study treatment will be summarized along with other disease characteristics.

### 5.3. Primary Efficacy Endpoint

All efficacy endpoints will be analyzed using the Full Analysis Set. The primary efficacy endpoint is objective response rate, defined as the proportion of participants with CR + PR. Tumor response and progression of cancer under study in real time will be evaluated locally at each study site according to RECIST v1.1.

To be assigned a status of PR or CR, changes in tumor measurements must be confirmed by repeat assessments that will be performed no less than 4 weeks after the criteria for response are first met. In order for a valid value of Stable Disease (SD) to be assigned, there must be evidence of stable disease for at least 7 weeks (the 8-week scan interval inclusive of a 1-week window per the SoA) from start of treatment. If the minimum time for SD has not been met on the first assessment, the assignment of BOR will depend on subsequent response assessments. Participants who do not have follow up data after a first assessment of SD prior to the minimum time requirement will be considered as not evaluable (NE).

The best overall response is determined by the following hierarchy: CR > PR > SD > PD > NE. Participants with a best overall response as confirmed CR or PR during the study will be



responders. Participants who had no post-baseline tumor assessment and those whose best overall response is no evaluable or less than CR or PR will be analyzed as non-responders.

### 5.3.1. Analysis of Objective Response Rate

The objective response rate and its 95% CI based on the Clopper-Pearson method will be provided. The proportion and 95% CI of participants with CR, PR, Stable Disease (SD), Progressive disease (PD) and Not Evaluable (NE) as defined by RECIST v1.1 will also be summarized and listed by visit.

Tumor size, defined as the sum of the target lesion diameters per RECIST v1.1, will be summarized as percent change from baseline by visit. In addition, the percent change from baseline in the sum of target lesion diameters as identified by RECIST v1.1 by the best overall response will be displayed graphically using a waterfall plot.

### 5.3.2. Sensitivity Analyses of Objective Response Rate

There is no sensitivity analysis of objective response rate. Post hoc analyses may be performed if deemed necessary.

# 5.3.3. Subgroup Analysis for Objective Response Rate

See Section 4.6 for subgroup analysis.

# 5.4. Secondary Efficacy Endpoints

Analysis of secondary endpoints will be conducted using the Full Analysis Set.

### 5.4.1. PFS-6

PFS-6 will be estimated using Kaplan-Meier method and 2-sided 95% CI based on log-log transformation. Participants who do not progress or die will be censored according to the censoring rules for the PFS as outlined in Table 3.

### 5.4.2. OS-2

The Kaplan-Meier method will be used to estimate the OS-2. Death due to any reasons will be an event. Participants who did not die at 2 years will be censored.



### 5.4.3. Change from Baseline in FOSI-8

Functional Assessment of Cancer Therapy (FACT) Ovarian Symptom Index-8 item version (FOSI-8) was used in this study for description of each item in FOSI-8 version 4, see Section 8.2.

Participants are asked to circle or make one number per statement to indicate their response as it applies to the past 7 days. In each statement, the numbers and meaning are as follows: 0 = Not at all, 1 = A little bit, 2 = Somewhat, 3 = Quite a bit, 4 = Very much. Except for statement 7 (I am content with the quality of my life right now), a lower number in the answer indicates a better condition. The response to the statements except for the statement 7 will be reversed and the sum of non-missing responses will be calculated.

The total FOSI-8 score will be summarized as sum of (8 question items) x 8 divided by the number of items answered. The FOSI-8 total score will range from 0 to 32 and a higher score is good. Therefore, a score of "0" is a severely symptomatic participant and the highest possible score is an asymptomatic participant. The FOSI-8 total score will be set to missing if 5 or more of the 8 item responses are missing.

Summary statistics of change from baseline in the FOSI-8 total score and the individual item responses will be summarized for each visit. In addition, the proportion of participants who achieved  $\geq 2$  improvement in FOSI-8 total score from baseline (Beaumont et al. 2007) will be summarized by each visit. Participants who could not possibly improve by at least 2 points due to a high score at baseline will be excluded from this analysis. A box and whisker plot displaying the total score over time by nominal visit and a figure for median change from baseline overtime will also be provided.

To evaluate association between changes of tumor size over time and the FOSI-8 total score, a figure with the percent change from baseline in tumor size on one y-axis and the change from baseline in FOSI-8 total score on a secondary y-axis over time (x-axis) will be generated.

# 5.4.4. Duration of Response (DoR)

DoR will be summarized with standard summary statistics and will also be analyzed using the Kaplan-Meier method for confirmed responders only. Quartiles (i.e., the 25th, 50th, and 75th percentile estimates) and the 2-sided 95% confidence intervals will be presented. If progression



or death was not observed, the participant will be censored according to the censoring rule for PFS (see Table 3). If there are censored participants in DoR, time to censoring will be used to summarize the range. The Kaplan-Meier plot will be provided.

By-participant listing will be provided for responders. The listing will include number of completed cycles before first response, date of first response, date of first disease progression or death if any, censored or event will be marked.

### 5.5. Exploratory Efficacy Endpoints

### 5.5.1. Time to Event Endpoints

Exploratory time to event endpoints include PFS, PFS on continued treatment, PFS2 and OS.

For each endpoint, quartiles (i.e., the 25th, 50th, and 75th percentile estimates) and the 2-sided 95% confidence intervals will be calculated from the Kaplan-Meier method. Survival probability and associated 95% CIs will be estimated at 6 months, 1 year, 18 months and 2 years as well. The number of events, number of participants censored, number of participants for each reason of censoring will be provided. The Kaplan-Meier plot of the survival distribution function will be presented with the number of participants at risk over time.

### **PFS**

For PFS, participants who have no documented disease progression and death will be censored according to the rules in Table 3. For PFS-6 and DoR, similar censoring rules should be used if applicable.

Table 3 PFS and DoR censoring rules

| Situation | Date of Censoring or Event | Outcome |
|---|---|---|
| No adequate tumor assessment at baseline or post-baseline and the participant has not died | Date of first dose of study treatment | Censored |
| No documented progression or death | Date of last adequate disease status assessment | Censored |



| Situation | Date of Censoring or Event | Outcome |
|---|---|---|
| Progression based on RECIST v1.1 with ≤1 missing consecutive scheduled tumor assessment before progression | Date of the earliest assessment that results in a finding of progression | Event |
| Death without documented progression with ≤1 missing consecutive scheduled tumor assessment before death | Date of death | Event |
| New anticancer therapy or procedure started prior to documented disease progression | Date of last adequate disease status assessment before the new therapy | Censored |
| Progression/Death after two or more missing scheduled tumor assessments | Date of last adequate disease status assessment before the missed assessments | Censored |

### Progression-free survival on continued nirogacestat treatment and PFS2

For the PFS analysis on continued nirogacestat treatment, only participants who continued the study treatment after the initial evidence of disease progression will be included. Participants who are alive and have not had a second progression will be censored at the last adequate disease status assessment date.

For PFS2, the second disease progression after participants discontinued the study treatment following the initial evidence of disease progression, and started the subsequent line of anticancer treatment, or death, whichever occurs first, will be considered as events for the PFS2 analysis. Participants who are alive and have not had a second progression on subsequent line of anticancer treatment will be censored at the last adequate disease status assessment date.

### OS

For OS, in participants who have died, death will be considered an event and the death date will be used to calculate the time. For participants who are alive at the time of analysis, who are lost to follow-up or who withdraw consent for follow-up, the OS endpoint will be censored on the last date that participants were known to be alive or lost to follow-up.



# 5.5.2. Next Generation Sequencing status

The NGS status will be assessed at baseline to detect FOXL2 C134W mutation as well as other genomic alterations and correlate these with response. A 2×2 table will be generated for FOXL2 C134W mutation (yes/no) vs. Objective Response (yes/no) to evaluate the correlation between mutation and ORR with the Spearman rank correlation and its 95% CI provided. Within each status, the percentage of participants with objective response (CR + PR) and its 2-sided exact 95% CI based on the Clopper-Pearson method will be provided. The response ratio of participants with alteration vs. those without alteration and its 95% CI will also be provided using the Farrington-Manning method.

NGS status data will be listed. Correlation between ORR and other genomic alterations will be analyzed post hoc if deemed necessary.

# 5.5.3. Inhibin A&B, Follicle-stimulating Hormone, Estradiol, CA-125, and AMH/Mullerian Inhibiting Substance (MIS)

Tumor and hormonal markers Inhibin A, Inhibin B, AMH/MIS, follicle-stimulating hormone, estradiol, and CA-125 will be assessed per the SoA (see Table 2 in the protocol). Summary statistics and change from baseline at each visit will be provided. Box and whisker plots displaying the values over time by nominal visit will also be provided.

To evaluate association between changes in tumor size over time with FSH and estradiol level, a figure with the percent change from baseline in tumor size on one y-axis and the change from baseline in FSH and estradiol level on a secondary y-axis over time (x-axis) will be generated.

# 5.5.4. Time to Response

Time to first objective response will be calculated as time in months from first dose until date of the first documented response (CR or PR). Only participants with confirmed response will be included and the time in months to first response will be summarized with standard summary statistics.

# 5.6. Safety Analyses

Safety analyses will be conducted using the Safety Analysis Set.



# 5.6.1. Study Dug Exposure and Compliance

Extent of exposure will be summarized as follows:

- Duration of exposure in months (last dose of study treatment date first dose date + 1 /30.4375) summarized as a continuous variable
- If a data cut-off date is used and some participants are receiving treatment at the time of analysis, the last dose date at the time of the data cut-off for analysis will be the data cut-off date
- Number and percentage of participants who received treatment with a duration of at least 1 cycle (28 days), 2 cycles, 3 cycles, 4 cycles, 5 cycles, 6 to 12 cycles, 13 to 25 cycles and 26 cycles or longer
- Actual dose intensity (mg/day) calculated as the cumulative dose received / duration of exposure in days
- Relative dose intensity (%) defined as 100 × (total cumulative dose received)/ (planned cumulative dose, where planned cumulative dose is 300 mg/day multiplied by duration of exposure in days) and summarized as a continuous variable
- Number and percentage of participants with a dose modification (dose reduction and/or dose interruption as reported on eCRF) as well as reasons for dose modification
- Number and percentage of participants with a dose reduction (as reported on eCRF)
- Time (in days) to the first dose reduction and first dose interruption will be summarized as continuous variables
- Number and percentage of participants with a dose interruption including the number of days interrupted
- Number and percentage of participants with study treatment discontinued
- Special Situations in exposure are defined as Abuse, Misuse, Occupational Exposure (inadvertent/accidental), or Medication Error of study treatment. The number and percentage of participants with each and overall special situations resulting in an adverse event will also be summarized.

A by-participant listing will be presented for exposure to study treatment and dosing modifications.



### 5.6.2. Adverse Events

All AEs will be coded using the MedDRA coding dictionary version 27.0 and displayed in tables and data listings using system organ class (SOC) and preferred term (PT).

Analyses of AEs will be performed for those events that are considered treatment-emergent adverse events (TEAEs), defined as those with initial onset or increasing in severity after the first dose of study treatment through 30 days after the last dose of study treatment. The imputation of partial/missing dates is described in Section 4.9.1.

Treatment-related TEAEs are defined as a TEAE that was considered by the Investigator to be related to the study treatment. If "Relationship to Study Treatment" is missing, it will be imputed as related in summary tables.

AE grade refers to the severity of the AE. The Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:

- Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated.
- Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting ageappropriate instrumental Activities of Daily Living (ADL).
- Grade 3 Severe or medically significant but not immediately life-threatening;
   hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL.
- Grade 4 Life-threatening consequences; urgent intervention indicated.
- Grade 5 Death related to AE.

An event is defined as 'serious' when it meets at least 1 of the predefined outcomes as described in the definition of an SAE (Protocol Appendix A5-1.3), not when it is rated as severe.

A summary of TEAEs will include the number and percentage of participants who experience at least one of the following. The total number of events will also be reported.

TEAEs



- TEAEs related to study treatment
- Serious TEAEs
- Serious TEAEs related to study treatment
- Serious TEAEs by maximum severity (Grade)
- TEAEs with CTCAE grade  $\geq 3$
- TEAEs with CTCAE grade  $\geq 3$  related to study treatment
- TEAEs by maximum severity (Grade)
- TEAEs leading to early discontinuation from study treatment
- TEAEs leading to early discontinuation from study treatment related to study treatment
- TEAEs leading to dose reduction
- TEAEs leading to dose reduction related to study treatment
- TEAEs leading to dose interruption
- TEAEs leading to dose interruption related to study treatment
- TEAEs leading to dose reduction or interruption
- TEAEs leading to dose reduction or interruption related to study treatment
- TEAEs leading to death
- TEAEs leading to death related to study treatment
- TEAEs by cycle of onset

In each tabulation of TEAEs, each participant will contribute only once (i.e., the most related occurrence, or the most intense occurrence, or the first cycle of onset) to each of the participant incidence rates in the descriptive analysis, regardless of the number of episodes.

The above categories will also be presented in tables summarizing SOC and PT, and sorted by descending frequency. If a participant experiences multiple AEs under the same PT (or SOC), the participant will be counted only once for that PT (or SOC). The number of events of each type will be displayed alongside associated participant incidence percentages.

A TEAE summary by PT only and sorted by descending frequency will also be produced.


All AEs will be listed in participant data listings. By-participant listings will also be provided for the following: TEAEs leading to death, serious adverse events, TEAEs leading to study treatment withdrawn, and TEAE leading to discontinuation from study.

# 5.6.3. Safety Topics of Special Interest

Safety topics of special interest have been identified based on review of safety data from prior studies with nirogacestat and include additional AEs beyond those specified in Protocol Section 11.3.1 as adverse events of special interest (AESIs). These safety topics of interest, including AESIs determined by the investigators for this study, will be summarized on separate tables. These safety topics, including AESIs, are defined for analysis purposes in different ways, including by using standardized MedDRA queries (SMQ) or customized MedDRA queries, and whether an investigator determined that an event was an AESI.

Unless specified otherwise, the incidence of AESIs based on the investigator's determination will be summarized by SOC and PT in tables and listed separately in participant data listings, and those by using defined lists of specific MedDRA PTs without regard to the investigator's designation of the reported event as an AESI will be summarized similarly.

For the safety topics of special interest (including AESIs) defined using standardized MedDRA queries (SMQ) or customized MedDRA queries, the specific MedDRA PTs for inclusion are all listed in Appendix 8.4 under the following groups. Safety topics for which narrow and broad terms are identified, only narrow terms are used for summary tables. The safety topics will be summarized by SOC and PT based on the Safety Analysis Set.

- Hypersensitivity
- Skin Disorder and Rash
- Hepatotoxicity
- Electrolyte Disorder
- Non-melanoma Skin Cancer
- Musculoskeletal Disorders
- Bone Fractures
- Mucositis/Stomatitis



- Hematologic Disorders
- Opportunistic Infections
- Central Nervous System Vascular Disorders
- Embolic and Thrombotic Events
- Cardiac Rhythm Disturbances
- Upper Respiratory Tract Infections
- Diarrhea

In addition to the summaries by SOC and PT as described above, separate summaries for concomitant medication use will be presented for the following safety topics:

- Hypophosphataemia (A subset of Electrolyte Disorder terms)
- Upper Respiratory Tract Infection
- Diarrhea
- Skin and Subcutaneous Rash (Broad and Narrow; a subset of Skin Disorder and Rash terms)
- Skin and Subcutaneous Rash (Narrow; a subset of Skin Disorder and Rash terms)

The number and percentage of participants with concomitant medication used for each safety topic of special interest will be presented by ATC Classification, Preferred Term and Grade (1-2 vs. ≥3). The following will be also summarized:

- Number and percentage of participants with the safety topic of special interest
- Time to Onset of First Instance of the safety topic of special interest (days)
- Duration of the safety topic of special interest (days) for each event
- Time from onset of first instance of the safety topic of special interest to resolution of last event
- Number of participants with the safety topic of special interest by outcome, grade (1-2 vs. ≥3), and dose modification (if any)
- Number and percentage of participants with concomitant medication use for the safety topic of special interest
- Duration of concomitant medication use for the safety topic of special interest (days)



If an adverse event is ongoing, the end date will be imputed as the data cut-off date for the duration calculation. The duration of concomitant medication use is defined as the number days a participant took medications for the safety topic of special interest. If multiple concomitant medications are taken on a given day, that day will be counted once in the sum. If a medication is ongoing, the end date will be imputed as the last visit date + 28 days (if not before the medication start date), or the study treatment end date if unavailable.

## 5.6.4. Protocol-Required Laboratory Assessments

Protocol-required laboratory parameters are listed in Table 13-1 in the protocol. The tests in this table will be performed by the local laboratory except for follicle-stimulating hormone (FSH), luteinizing hormone (LH), estradiol, progesterone, Inhibin A, Inhibin B, Anti-Mullerian hormone/Mullerian inhibiting substance (AMH/MIS), and CA-125, which will be sent to a central laboratory.

Clinical laboratory values will be expressed in international system of units (SI) units. Summaries of clinical laboratory parameters will be summarized by study visit and overall. Tables for the shift of laboratory data from baseline to the worst post-baseline value will be presented for each lab parameter. The shift from baseline to each visit will also be presented for hematology and chemistry parameters.

The actual value and change from baseline will be summarized for each visit for clinical hematology and chemistry. For analysis of tumor markers and hormones, see Section 5.5.3.

Laboratory results will also be summarized by maximum CTCAE grade as available. For lab tests with NCI – CTCAE classification, the shift from baseline to each post baseline visit and the maximum (worst) post baseline grade will be tabulated. Shift tables will summarize the count and frequency of each baseline CTCAE grade to the highest CTCAE grade on study. Laboratory tests with bi-directional grades will be presented separately for each direction (e.g., hyperglycemia and hypoglycemia). For lab tests without NCI – CTCAE classifications, the shift from baseline to each post baseline visit and the worst post-baseline value (high or low) will be summarized using the lab range indicators (normal, high, or low).



Additional shift tables will be produced for ALT, AST, alkaline phosphatase, bilirubin, phosphorus, and creatine showing shifts of below normal range, within normal range, >1 to  $2 \times 10^{-5}$  upper limit of normal range, >2 to  $3 \times 10^{-5}$  upper limit of normal range, >3 to  $5 \times 10^{-5}$  upper limit of normal range from baseline to the worst (highest) post baseline value.

Box and whisker plots displaying the values over time by nominal visit will be produced for the hematology and clinical chemistry lab tests.

All laboratory results will be listed and laboratory tests with an abnormal result will be flagged. A subset listing will be presented for all grade 3 or higher laboratory values.

A summary table and a listing of participants meeting liver chemistry stopping criteria will be provided by the cycle of onset and overall. These are participants with the following conditions:

- ALT  $>5 \times ULN$
- ALT  $\geq 3 \times ULN$  persists for  $\geq 4$  weeks
- ALT  $\ge 3 \times ULN$  and bilirubin  $\ge 2 \times ULN$  (> 35% direct bilirubin)
- ALT  $\ge 3 \times \text{ULN}$  and International normalized ratio (INR) > 1.5, if INR measured
- ALT ≥ 3×ULN and cannot be monitored weekly for 4 weeks. Missing lab values within window will be considered not monitored.
- ALT ≥ 3×ULN associated with symptoms (new or worsening) believed to be related to liver

Serum pregnancy testing data will be presented for each participant in a data listing.

# 5.6.5. Physical Exam and Eastern Cooperative Oncology Group Performance Status

Physical examination abnormalities reported as AEs will be summarized along with other TEAEs.

Shift tables will be used to summarize the count and frequency for each shift of baseline ECOG performance status grade to the worst and the best post-baseline ECOG grade. The ECOG performance status grades are outlined in Table 4.



All physical examination findings and ECOG performance status results will be presented in data listings.

**Table 4 Eastern Cooperative Oncology Group Performance Status Grades** 

| Grade | Description |
|---|---|
| 0 | Normal activity. Fully active, able to carry on all pre-disease performance without restriction. |
| 1 | Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work). |
| 2 | In bed < 50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours. |
| 3 | In bed > 50% of the time. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. |
| 4 | 100% bedridden. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair. |
| 5 | Dead. |

Source: Oken MM, Creech RH, Tormey DC, et al. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982; 5:649-655

# 5.6.6. Electrocardiogram

The actual value and change from baseline at each time point will be summarized for 12-lead ECG parameters. The 12-Lead ECG parameters include heart rate, PR, RR, QRS, QT and QTcF intervals.

Categorical groups of QTcF will be summarized as follows:

- Maximum post-baseline QTcF
  - $\circ \le 450 \text{ msec}$
  - $\circ$  > 450 and  $\leq$  480 msec
  - $\circ$  > 480 and  $\leq$  500 msec
  - $\circ$  > 500 msec



- Maximum change from baseline for QTcF
  - o < 30 msec
  - $\circ$  > 30 and  $\leq$  60 msec
  - $\circ$  > 60 msec
- Baseline QTcF < 450 msec and post-baseline QTcF > 500 msec
- Baseline QTcF between 450 and 480 msec and post-baseline QTcF ≥ 530 msec

ECG parameters will be summarized by visit and the worst post-baseline change from baseline. All ECG data will be included in a by-participant data listing. Listings will be provided for participants with abnormal or outlying values for QTcF and changes in QTcF.

# 5.6.7. Vital Signs

The actual value and change from baseline for all parameters (blood pressure, respiratory rate, heart rate, and body temperature) will be summarized at each scheduled visit.

Potentially clinically significant post-baseline vital signs will also be summarized following the criteria as below:

- Systolic Blood Pressure (mmHg)
  - Value  $\geq 150$
  - Increase of 20 from baseline
  - O Value  $\geq 150$  and increase of 20 from baseline
  - Value < 90
  - Decrease of 20 from baseline
  - Value < 90 and decrease of 20 from baseline
- Diastolic Blood Pressure (mmHg)
  - Value  $\geq$  95
  - Increase of 10 from baseline
  - Value  $\ge$  95 and increase of 10 from baseline
  - $\circ$  Value < 60
  - Decrease of 10 from baseline
  - Value < 60 and decrease of 10 from baseline



- Heart Rate (beats/min)
  - Value  $\geq 110$
  - o Increase of 20 from baseline
  - Value  $\ge 110$  and increase of 20 from baseline
  - $\circ$  Value < 50
  - o Decrease of 20 from baseline
  - Value  $\leq$  50 and decrease of 20 from baseline
- Temperature (°C)
  - Value  $\geq 38$
  - o Value < 35

Vital sign measurements will be summarized by visit and the worst post-baseline change from baseline. The data listing will be presented for each participant. A summary table and listing will also be provided for participants with potentially clinically significant vital signs.

#### 5.6.8. Concomitant Medications

Any medication or vaccine (including over-the-counter or prescription medicines, vitamins, and/or herbal supplements) that the participant is receiving at the time of informed consent and/or receives during the study through 30 days after the last dose of study treatment will be recorded along with:

- Reason for use;
- Dates of administration including start and end dates; and
- Dosage information including dose and frequency.

Concomitant medications will be coded using the WHO Drug Dictionary March 2022 version or higher. Medications or vaccines that ended before receiving the first study treatment will be considered as the prior medication. Medications or vaccines that continued or started on or after receiving the first dose through 30 days after the last dose of study treatment will be summarized as the concomitant medication. Medication, vaccine or procedure started more than 30 days after the last dose will be considered as subsequent.



The handling of partial/missing start dates for concomitant therapies/medications are described in Section 4.9.2. Concomitant medications will be tabulated by anatomic therapeutic class (ATC) and PT. In these tabulations, each participant will contribute only once to each ATC and PT regardless of number of uses.

The concomitant procedures will be coded using the MedDRA coding dictionary version 27.0 and displayed in tables and data listings using system organ class (SOC) and preferred term (PT).

All medications, vaccines and procedures will be included in data listings. An identifier will be used to show whether a medication, vaccine or procedure was prior, concomitant or subsequent.

# 5.7. Pharmacokinetic and Pharmacodynamic Analyses

Exploratory analyses maybe conducted based on the data collected, with purposes of providing information for potential pharmacokinetic/pharmacodynamic (PK/PD) analysis if deemed necessary. The specifics of these analyses will be described in a separate PK/PD Analysis Plan and reported separately from the main Clinical Study Report (CSR). For purposes of the CSR for which this SAP provides the basis, serum pharmacokinetic collection dates, times, and concentrations will be displayed in a data listing. Additionally, summaries of the concentrations will be provided.

# 5.8. Interim Analysis

No formal interim analysis is planned. This study planned to use a Bayesian approach of continuous monitoring for early futility stopping based on ORR Potential timepoints for interim evaluation might occur when 10, 20, and 30 participants had completed 6 months of follow-up or dropped out. At each interim look, an exact 2-sided 95% CI based on the Clopper-Pearson method would also be provided. See Section 1.4 for a brief description of both methods.

This section provides detailed calculation of the Bayesian approach, however, due to the rapid enrollment, the previously planned informal data assessment using this Bayesian approach for early futility stopping based on ORR was no longer feasible as instead of 10 participants, 53 were already enrolled before the one year predicted cutoff time point.



The Bayesian approach to be used for futility analysis assumes a beta-binomial distribution with an uninformative prior of beta distribution. If a random variable Z follows a beta distribution with parameters  $(\alpha, \beta)$ , the probability density function will be

(1) 
$$f(z) = \frac{z^{\alpha-1}(1-z)^{\beta-1}}{B(\alpha,\beta)},$$

where potential values of z are in (0,1),

(2) 
$$B(\alpha, \beta) = \Gamma(\alpha)\Gamma(\beta)/\Gamma(\alpha, \beta),$$

and  $\Gamma$  is the Gamma function, i.e.,  $\Gamma(\alpha) = \int_0^\infty t^{\alpha-1} e^{-t} dt$ . The mean of Z is  $\alpha/(\alpha+\beta)$ .

At the first interim look, the prior of ORR is assumed to follow a beta distribution with parameter (0.1, 0.9). Hence the corresponding mean is 0.1. Assume at an assessment point, the study has accrued X responders out of n (<43) participants. With a prior distribution of beta (a, b), X follows a binomial distribution and the posterior distribution of the response rate follows a beta distribution with parameters (a+x, b+n-x), where x is the observed value of X (Lee and Liu 2008; Chen et al. 2019). For example, if 2 out of 10 participants are responders at the first interim look, the updated prior of ORR will follow a beta distribution with parameters (2.1, 8.9), which has a mean of 2.1/11=19.1%. Hence, the initially assumed beta prior with parameters (0.1, 0.9) does not have substantial impact on the updated prior and is considered non-informative prior.

For the remaining (43-n) future participants, the number of responses, Y, follows a beta-binomial distribution with parameters (43-n, a+x, b+n-x) (Lee and Liu 2008). Since a, b, n, x are known at this point, the probability Pr(Y=i) can be calculated using the probability mass function of a beta-binomial distribution. See equation (3) below.

If Z follows a beta-binomial distribution with parameters (n, a, b), the probability of Z = z is:

(3) 
$$f(z|n,a,b) = \binom{n}{z} \frac{B(z+a,n-z+b)}{B(a,b)}$$

If *i* out of (43-n) future participants are responders, the updated prior for ORR will follow a beta distribution with parameters (0.1+x+i, 0.9-x-i). If under the frequentist framework, the null hypothesis is ORR =15%. the posterior probability of ORR >15% can be calculated. Using SAS® CDF function, this probability is:



(4) 
$$pr(ORR > 0.15|x, Y = i) = 1 - CDF("Beta", 0.15, (0.1 + x + i), (0.9+43-x-i)).$$

Define the predictive probability as the chance of observing any Y = i responders in future participants such that the posterior probability of ORR >0.15 is greater than 85%. If the predictive probability is too low, e.g.,  $\leq 10\%$ , the study may be terminated for futility.

From the observed responders x and a target ORR, the predictive probability of reaching the target ORR at the end of study can be calculated with the beta-binomial distribution as follows. After observing a total of x out of n responders up to an interim look, the possible number of responders, Y, in the future will be 0, 1, 2, ..., (43-n). For each possible Y = i, calculate the posterior probability of  $Pr_i(ORR > 0.15|x, Y=i)$ , where i=0, i=0, i=0, i=0, ..., i=0, using equation (4). If this posterior probability is i=0.85, i=0 responders is considered promising. The probability of i=0 can be calculated using equation (3). The predictive probability for ORR i=0 with threshold 85% is:

(5) *Predictive probability* 

$$= \sum_{i=0}^{43-n} \{ \operatorname{pr}(Y = i | x) \times I[\operatorname{pr}(ORR > 0.15 | x, Y = i) > 0.85] \},$$

where pr(Y = i|x) is the probability of observing i responders in future (43-n) participants given x out of n responders, and I[pr(ORR > 0.15|x, Y = i) > 0.85]=1 if the statement inside [] is true; otherwise, the value of I is 0. In summary, the predictive probability in equation (5) can be calculated using the following algorithm:

- 1) Assign predictive probability pp to 0.
- 2) For i=0 to 43-n,
  - a. Calculate the posterior probability ps = pr(ORR > 0.15 | x, Y = i) using equation (4).
  - b. If ps > 0.85, do the following:
    - i. Calculate the probability of observing Y = i conditional on observing x responders using the beta-binomial distribution with parameters (43-n, x+0.1, n-x+0.9), i.e.,

(6) 
$$\Pr(Y = i|x)$$



$$= {43 - n \choose i} \frac{B(i + x + 0.1, 43 - n - i + n - x + 0.9)}{B(a, b)}$$
$$= {43 - n \choose i} \frac{B(i + x + 0.1, 43 - i - x + 0.9)}{B(x + 0.1, n - x + 0.9)}.$$

- ii. Update predictive probability pp with pp+pr(Y = i|x).
- c. After completing the loop in 2), the final *pp* is the predictive probability of ORR >0.15 with threshold 0.85.

In addition to using the Bayesian approach to calculate the predictive probability of observing a promising ORR, the frequentist approach will also be applied by generating the exact 95% CI of ORR based on the Clopper-Pearson method.

To evaluate the robustness of the observed result, the number of observed responders will be decreased and increased by 1, 2, and 3 (as long as the resulting ORR is between 0 and 100%) to repeat the analyses of ORR.



#### 6. CHANGES TO PLANNED ANALYSES

Notable changes from the protocol-defined statistical analyses compared to this statistical analysis plan are described below:

- I. PFS-6 was redefined as a survival probability.
- II. Definitions and analysis method were added for PFS and OS.
- III. The planned informal interim analysis using the Bayesian approach for early futility stopping based on ORR was not performed. Due to this study's rapid enrollment, it was not feasible to perform the planned informal interim analysis using the Bayesian approach because, instead of 10 participants, 53 were enrolled before the one year predicted cutoff time point.
- IV. Additional preferred terms were added in electrolyte abnormalities protocol Section
   4.3 vs. SAP section 8.4.1.4.



#### 7. REFERENCES

Brown, J., W.E. Brady, J. Schink, L. Le, M. Leitao, S. D. Yamada, K. Geest, and D.M. Gershenson. 2014. "Efficacy and Safety of Bevacizumab in Recurrent Sex Cord-stromal Ovarian Tumors: Results of a Phase 2 Trial of the Gynecologic Oncology Group." Cancer 120 (3): 344–51. https://doi.org/10.1002/cncr.28421.

Chen, D-T., M.J. Schell, W.J. Fulp, F. Pettersson, S. Kim, J.E. Gray, and E.B. Haura. 2019. "Application of Bayesian Predictive Probability for Interim Futility Analysis in Single-Arm Phase II Trial." Translational Cancer Research 8 (Suppl 4): S404–20. https://doi.org/10.21037/tcr.2019.05.17.

Eisenhaur EA, Therasse P, et al. New response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan; 45(2):228-47.

European Medicines Agency. Guidance on the Management of Clinical Trials During the COVID-19 (Coronavirus) Pandemic. 2021 April 02 (Version 4.0).

Farrington CP, Manning G. Test statistics and sample size formulae for comparative binomial trials with null hypothesis of non-zero risk difference or non-unity relative risk. Statist. Med. 1990;9(12):1447–1454.

Lee, J., and D. Liu. 2008. "A Predictive Probability Design for Phase II Cancer Clinical Trials." Clinical Trials 5 (2): 93–106. <a href="https://doi.org/10.1177/1740774508089279">https://doi.org/10.1177/1740774508089279</a>.

Oken MM, Creech RH, Tormey DC, et al. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982; 5:649-655.

Ray-Coquard, I., P. Harter, D. Lorusso, C. Dalban, I. Vergote, K. Fujiwara, L. Gladieff, et al. 2020. "Effect of Weekly Paclitaxel With or Without Bevacizumab on Progression-Free Rate Among Patients With Relapsed Ovarian Sex Cord-Stromal Tumors." JAMA



Oncology 6 (12): 1923–30. https://doi.org/10.1001/jamaoncol.2020.4574.

US Food and Drug Administration. Conduct of Clinical Trials of Medical Products During the COVID-19 Public Health Emergency. Guidance for Industry, Investigators, and Institutional Review Boards. March 2020 (Updated Jan 2021).

J. Beaumont, S. Yount, D. Lalla, D. Lubeck, M. Derynck, B. Karlan, and D. Cella. 2007. "Validation of the Functional Assessment of Cancer Therapy-Ovarian (FACT-O) Symptom Index (FOSI) in a Phase II Clinical Trial of Pertuzumab in Patients with Advanced Ovarian Cancer". Journal of Clinical Oncology 25 (18\_suppl). https://doi.org/10.1200/jco.2007.25.18\_suppl.160.



#### 8. APPENDICES

#### 8.1. RECIST Criteria V1.1

For full guidelines, see RECIST Criteria v1.1 (Eisenhauer 2009).

#### **Categorizing lesions at Baseline:**

• Only participants with measurable disease (i.e., at least one measurable lesion) at screening are included.

Measurable lesion – Lesion that can be accurately measured in at least one dimension (longest diameter [LD]) in the plane of measurement is to be recorded) and with longest diameter at least twice the slice thickness and at least 10 mm when assessed by computed tomography (CT) or magnetic resonance imaging (MRI)

- Measurable disease will be assessed by CT or MRI.
- The same method of assessment (CT or MRI) and the same technique will be used to characterize each identified and reported lesion at screening and during follow-up.
- Target Lesions up to 2 lesions per organ and 5 lesions in total, representative of all involved organs at Baseline.
- Non-target Lesion-All other lesions (or sites of disease) will be identified as non-target lesions and should also be recorded at baseline. Measurements of these lesions are not required, but the presence or absence of each should be noted throughout follow-up.

#### **Methods of Measurement**

CT or MRI must be used to measure target lesions selected for response assessment.

Conventional CT and MRI will be performed with cuts of 10 mm or less in slice thickness contiguously.

# **Recording Tumor Assessments**

All sites of disease must be assessed at screening. Screening assessment must be done within 28 days of starting study treatment. For an adequate screening assessment, all required scans must be done within 28 days prior to first dose of study treatment and all disease must be documented appropriately.



At follow-up, disease site must be assessed using the method (CT or MRI) and same technique as screening, including consistent administration of contrast (CT only) and timing of scanning. If a change needs to be made the case must be discussed with the Sponsor.

Unequivocal new lesions will be recorded at follow-up time points. Measurement of new lesions is not required. If a new lesion is equivocal, for example because of its small size, continued therapy and follow-up evaluation will clarify if it represents truly new disease. If repeat scans confirm there is definitely a new lesion, then progression should be declared using the date of the initial scan.

## Response Criteria: Evaluation of target lesions

| Complete Response (CR): | Disappearance of all target lesions. |
|---|---|
| Partial Response (PR): | At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum of LD. |
| Progressive Disease (PD): | At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum of LD recorded since the treatment started or the appearance of one or more unequivocal new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. |
| Stable Disease (SD): | Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started. |

## **Evaluation of best overall response**

The best overall response is the best response recorded from the start of the study treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the start of study treatment). The participant's best response assignment will depend on the achievement of both measurement and confirmation criteria (defined below).



#### Time point response: participants with target disease

| <b>Target Lesions</b> | Nontarget Lesions | New Lesions | <b>Overall Response</b> |
|---|---|---|---|
| CR | CR | No | CR |
| CR | Non-CR/non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or not all evaluated | No | PR |
| SD | Non-PD or not all evaluated | No | SD |
| Not all evaluated | Non-PD | No | NE |
| PD | Any | Yes or No | PD |
| Any | PD | Yes or No | PD |
| Any | Any | Yes | PD |

CR=Complete Response; NE=Not Evaluable; PD=Progressive Disease; PR=Partial Response; SD=Stable Disease.

Participants with a global deterioration of health status requiring discontinuation of study treatment without objective evidence of disease progression at that time will be classified as having "symptomatic deterioration". Every effort should be made to document the objective progression even after discontinuation of treatment.

#### Confirmation

#### • Confirmation of response:

- The main goal of confirmation of objective response is to avoid overestimating the response rate observed. In cases where confirmation of response is not feasible, it should be made clear when reporting the outcome of such studies that the responses are not confirmed.
- To be assigned a status of PR or CR, changes in tumor measurements must be confirmed by repeat assessments that will be performed no less than 4 weeks after the criteria for response are first met.
- Confirmation of SD: in the case of SD, follow-up measurements must have met the SD criteria at least once after study entry (signing of Informed Consent Form [ICF]) at a minimum interval of 8 weeks.

#### **Duration of overall response**

• The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever status is recorded first) until the first date that recurrence



or PD is objectively documented, taking as reference for PD the smallest measurements recorded since the treatment started.

#### **Duration of stable disease**

• SD is measured from the start of the treatment until the criteria for disease progression are met, taking as reference the smallest measurements recorded since the treatment started.



# 8.2. FACT/NCCN Ovarian Symptom Index (FOSI) - Version 4

Below is a list of statements that other people with your illness have said are important. Please circle or mark one number per line to indicate your response as it applies to the <u>past 7</u> days.

| | | Not at<br>all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|
| G | I have a lack of energy | 0 | 1 | 2 | 3 | 4 |
| C | I have been vomiting | 0 | 1 | 2 | 3 | 4 |
| G | I have pain | 0 | 1 | 2 | 3 | 4 |
| G | I have nausea | 0 | 1 | 2 | 3 | 4 |
| ( | I have swelling in my stomach area | 0 | 1 | 2 | 3 | 4 |
| G | I worry that my condition will get worse | 0 | 1 | 2 | 3 | 4 |
| G | I am content with the quality of my life right | 0 | 1 | 2 | 3 | 4 |
| | I have cramps in my stomach area | 0 | 1 | 2 | 3 | 4 |
| C | | | | | | |

#### Instructions:\*

- 1. Record answers in "item response" column. If missing, mark with an X
- 2. Perform reversals as indicated, and sum individual items to obtain a score.
- 3. Multiply the sum of the item scores by the number of items in the subscale, then divide by the number of items answered. This produces the symptom index score.
- 4. As with all FACIT questionnaires, a high score is good. Therefore, a score of "0" is a severely symptomatic patient and the highest possible score is an asymptomatic patient.

Divide by number of items answered:

| <u>Subscale</u> | <u>Item Code</u> | Reverse item | ? | <u>Item response</u> | <u>Item Score</u> |
|---|---|---|---|---|---|
| FOSI | GP1 | 4 | - | | = |
| | 02 | 4 | - | | = |
| | GP4 | 4 | - | | = |
| Score range: 0-32 | GP2 | 4 | - | | = |
| | 01 | 4 | - | | = |
| | GE6 | 4 | - | | = |
| | GF7 | 0 | + | | = |
| | 03 | 4 | - | | = |
| | | | | Sum individual item scores:<br>Multiply by 8: | |

Page 55 of 100



# 8.3. Mock-up Tables, Listings, and Figure

Mock-up tables, listings and figures are in separate documents.

# 8.4. Safety Topics of Special Interest Preferred Terms

This appendix outlines the definition of treatment-emergent AESIs. Additional attention will specifically be given to the safety topics of special interest identified using SMQ or customized MedDRA queries based on MedDRA version 27.0.

# 8.4.1. Protocol-Specified AESIs

Ovarian Toxicity is specified in the protocol as an AESI. However, the majority of participants in this study will not menstruate since they have had their ovaries or uteruses, or both, surgically removed, or were documented to be post-menopausal. Therefore, it will not be relevant to assess ovarian toxicity in this study so the Preferred Terms defining Ovarian Toxicity are not included in this section.

# 8.4.1.1. Hypersensitivity

The Hypersensitivity search definition is a custom MedDRA version 27.0 query based on selected terms from the Anaphylactic reaction SMQ, Angioedema SMQ, and Allergic conditions High Level Group Term (HLGT). The PTs are listed below, and all will be considered Narrow search terms:

Acquired C1 inhibitor deficiency Laryngotracheal oedema

AGEP-DRESS overlap Limbal swelling

Allergic oedema Lip oedema

Allergic reaction to excipient Lip swelling

Anaphylactic reaction Mouth swelling

Anaphylactic shock Multiple drug hypersensitivity

Anaphylactic transfusion reaction Oculorespiratory syndrome

Anaphylactoid reaction Oedema mouth

Anaphylactoid shock Orbital oedema



Angioedema Orbital swelling

Circulatory collapse Oropharyngeal oedema

Circumoral oedema Oropharyngeal swelling

Circumoral swelling Palatal oedema

Conjunctival oedema Palatal swelling

Corneal oedema Periorbital oedema

Dermatitis allergic Periorbital swelling

Dialysis membrane reaction Pharyngeal oedema

Drug eruption Pharyngeal swelling

Drug hypersensitivity Procedural shock

Drug reaction with eosinophilia and systemic symptoms Scleral oedema

Epiglottic oedema Severe cutaneous adverse reaction

Erythema multiforme Shock

Eye oedema Shock symptom

Eye swelling SJS-TEN overlap

Eyelid oedema Stevens-Johnson syndrome

Face oedema Swelling face

Fixed eruption Swelling of eyelid

Gingival oedema Swollen tongue

Gingival swelling Systemic contact dermatitis

Gleich's syndrome Tongue oedema

Hereditary angioedema Toxic epidermal necrolysis

Hereditary angioedema with C1 esterase inhibitor

deficiency Toxic skin eruption

Hereditary angioedema with normal C1 esterase inhibitor Tracheal oedema

Hypersensitivity Type I hypersensitivity

Idiopathic angioedema Type II hypersensitivity



Type III immune complex Idiopathic histaminergic angioedema mediated reaction

Idiopathic urticaria Type IV hypersensitivity reaction

Intestinal angioedema Urticaria

Kounis syndrome Urticaria cholinergic

Laryngeal oedema Urticaria chronic

Urticaria papular

#### 8.4.1.2. Skin Disorder and Rash

The Skin Disorder and Rash search definition is a custom MedDRA version 27.0 query based on selected terms from the Skin and subcutaneous tissue disorders and Infections and infestations System Organ Classes (SOCs). Analyses of skin disorders will be presented for both narrow and broad terms. It is grouped into hidradenitis, skin and subcutaneous rash, and hair follicle subcategories. The PTs are listed below, with Narrow search terms indicated:

#### **Hidradenitis:**

Hidradenitis<sup>1</sup>

Sweat gland infection

Abscess sweat gland

Groin sinus excision

Groin abscess

#### Skin and subcutaneous rash:

Acne Rash erythematous<sup>1</sup>

Acne conglobata Rash follicular<sup>1</sup>

Acne cystic Rash macular<sup>1</sup>

Acne pustular Rash maculo-papular<sup>1</sup>

Dermatitis acneiform Rash maculovesicular

<sup>&</sup>lt;sup>1</sup> Narrow term.



Dermatitis exfoliative Rash morbilliform<sup>1</sup>

Dermatitis exfoliative generalised Rash papular<sup>1</sup>

Dermatitis<sup>1</sup> Rash papulosquamous<sup>1</sup>

Dry skin Rash pruritic<sup>1</sup>

Erythema<sup>1</sup> Rash pustular

Erythrodermic atopic dermatitis Rash rubelliform

Exfoliative rash Rash scarlatiniform

Mucocutaneous rash Rash vesicular

Nodular rash<sup>1</sup> Rash<sup>1</sup>

Pruritus Skin exfoliation

Pustule Vasculitic rash

#### Hair Follicle:

Abscess of eyelid Eyelid infection

Acne Follicular disorder

Acne conglobata Folliculitis<sup>1</sup>

Acne cosmetica Folliculitis barbae

Acne cystic Folliculitis genital

Acne fulminans Furuncle<sup>1</sup>

Acne infantile Hordeolum

Acne occupational Oil acne

Acne varioliformis Pyoderma

Alopecia areata<sup>1</sup> Pyoderma streptococcal

Alopecia totalis<sup>1</sup> Rash pustular<sup>1</sup>

Alopecia universalis<sup>1</sup> Skin bacterial infection

Alopecia<sup>1</sup> Staphylococcal skin infection

Carbuncle Subcutaneous abscess

<sup>&</sup>lt;sup>1</sup> Narrow term.



Dermatitis acneiform

Diffuse alopecia<sup>1</sup>

Eyelid boil

Eyelid folliculitis

# 8.4.1.3. Hepatotoxicitiy

The Hepatotoxicity search definition is a custom MedDRA version 27.0 query based on Narrow and Broad terms from the Drug related hepatic disorders - comprehensive search SMQ, Cholestasis and jaundice of hepatic origins SMQ, Drug related hepatic disorders SMQ– severe events only, Liver related investigations, signs and symptoms SMQ, and Liver related coagulation and bleeding disturbances SMQ. The PTs are listed below, with Narrow search terms indicated:

5'nucleotidase increased Hepatic hypoperfusion

Acquired antithrombin III deficiency Hepatic lymphocytic infiltration

Acquired factor IX deficiency Hepatic mass

Acquired factor V deficiency<sup>1</sup> Hepatic pain

Acquired factor VIII deficiency Hepatic sequestration

Acquired factor XI deficiency Hepatic vascular resistance increased

Acquired hepatocerebral degeneration Hepatic venous pressure gradient abnormal

Acquired protein S deficiency Hepatic venous pressure gradient increased

Acute graft versus host disease in liver Hepatobiliary cancer

Acute hepatic failure<sup>1</sup> Hepatobiliary cancer in situ

Acute on chronic liver failure Hepatobiliary cyst

Acute yellow liver atrophy Hepatobiliary disease

Alanine aminotransferase abnormal<sup>1</sup> Hepatobiliary neoplasm

Alanine aminotransferase increased<sup>1</sup> Hepatobiliary scan abnormal

<sup>&</sup>lt;sup>1</sup>Narrow term.



Allergic hepatitis Hepatoblastoma

Alloimmune hepatitis Hepatoblastoma recurrent

Ammonia abnormal Hepatocellular carcinoma

Ammonia increased Hepatocellular foamy cell syndrome

Anorectal varices Hepatocellular injury

Anorectal varices haemorrhage Hepatomegaly

Anti factor X activity abnormal Hepatopulmonary syndrome

Anti factor X activity decreased Hepatorenal failure

Anti factor X activity increased Hepatorenal syndrome

Anti-liver cytosol antibody type 1 positive<sup>1</sup> Hepatosplenomegaly

Antithrombin III decreased Hepatotoxicity<sup>1</sup>

Ascites Hyperammonaemia

Aspartate aminotransferase abnormal<sup>1</sup> Hyperbilirubinaemia

Aspartate aminotransferase increased<sup>1</sup> Hypercholia

AST to platelet ratio index increased Hyperfibrinolysis

AST/ALT ratio abnormal Hypertransaminasaemia

Asterixis Hypoalbuminaemia

Autoimmune hepatitis Hypocoagulable state

Bacterascites Hypofibrinogenaemia

Benign hepatic neoplasm Hypoprothrombinaemia

Benign hepatobiliary neoplasm Hypothrombinaemia

Bile acids abnormal<sup>1</sup> Hypothromboplastinaemia

Bile acids increased Icterus index increased

Bile output abnormal Immune-mediated cholangitis

Bile output decreased Immune-mediated hepatic disorder

Biliary ascites Immune-mediated hepatitis

Biliary cirrhosis Increased liver stiffness



Biliary fibrosis International normalised ratio abnormal

Bilirubin conjugated abnormal International normalised ratio increased

Bilirubin conjugated increased Intestinal varices

Bilirubin excretion disorder Intestinal varices haemorrhage

Bilirubin urine present Intrahepatic portal hepatic venous fistula

Biopsy liver abnormal Ischaemic hepatitis

Blood alkaline phosphatase abnormal Jaundice

Blood alkaline phosphatase increased Jaundice cholestatic

Blood bilirubin abnormal Jaundice hepatocellular

Blood bilirubin increased Kayser-Fleischer ring

Blood bilirubin unconjugated increased Leucine aminopeptidase increased

Blood cholinesterase abnormal Liver and pancreas transplant rejection

Blood cholinesterase decreased Mixed liver injury

Blood fibrinogen abnormal Ocular icterus

Blood fibringen decreased Parenteral nutrition associated liver disease

Blood thrombin abnormal Liver carcinoma ruptured

Blood thrombin decreased Liver dialysis

Blood thromboplastin abnormal Liver disorder

Blood thromboplastin decreased Liver injury

Bromosulphthalein test abnormal Liver-kidney microsomal antibody positive<sup>1</sup>

Cardiohepatic syndrome Liver operation

Child-Pugh-Turcotte score abnormal Liver sarcoidosis

Child-Pugh-Turcotte score increased Liver transplant

Cholaemia Liver transplant failure

Cholangiosarcoma Liver transplant rejection

Cholestasis Lupoid hepatic cirrhosis

Cholestatic liver injury Lupus hepatitis



Cholestatic pruritus Mixed hepatocellular cholangiocarcinoma

Chronic graft versus host disease in liver Multivisceral transplantation

Chronic hepatic failure Nodular regenerative hyperplasia

Chronic hepatitis Nonalcoholic fatty liver disease

Coagulation factor decreased Non-alcoholic steatohepatitis

Coagulation factor IX level abnormal Non-cirrhotic portal hypertension

Coagulation factor IX level decreased Oedema due to hepatic disease

Coagulation factor V level abnormal Oesophageal varices haemorrhage

Coagulation factor V level decreased Peripancreatic varices

Coagulation factor VII level abnormal Peritoneovenous shunt

Coagulation factor VII level decreased Portal fibrosis

Coagulation factor X level abnormal Portal hypertension

Coagulation factor X level decreased Portal hypertensive colopathy

Coma hepatic Portal hypertensive enteropathy

Complications of transplanted liver Portal hypertensive gastropathy

Computerised tomogram liver abnormal Portal shunt

Congestive hepatopathy Portal shunt procedure

Cryptogenic cirrhosis Portal tract inflammation

Cytokeratin 18 increased Portal vein cavernous transformation

Deficiency of bile secretion Portal vein dilatation

Diabetic hepatopathy Portopulmonary hypertension

Drug-induced liver injury Primary biliary cholangitis

Duodenal varices Radiation hepatitis

Factor VII activity decreased<sup>1</sup>

Flood syndrome Regenerative siderotic hepatic nodule

Focal nodular hyperplasia Renal and liver transplant

Foetor hepaticus Retrograde portal vein flow



Galactose elimination capacity test abnormal

Galactose elimination capacity test decreased

Gallbladder varices

Gamma-glutamyltransferase abnormal<sup>1</sup>

Gamma-glutamyltransferase increased<sup>1</sup>

Gastric variceal injection

Gastric variceal ligation

Gastric varices

Gastric varices haemorrhage

Gastrooesophageal variceal haemorrhage

prophylaxis

Glutamate dehydrogenase increased

Glycocholic acid increased

Graft versus host disease in liver

Granulomatous liver disease

Hepatitis cholestatic

Haemangioma of liver

Haemorrhagic hepatic cyst

Hepatectomy

Hepatic adenoma

Hepatic angiosarcoma

Hepatic atrophy

Hepatic calcification

Hepatic cancer

Hepatic cancer metastatic

Hepatic cancer recurrent

Hepatic cancer stage I

Reye's syndrome

Reynold's syndrome

Small-for-size liver syndrome

Spider naevus

Splenic artery embolisation

Splenic varices

Splenic varices haemorrhage

Splenorenal shunt

Splenorenal shunt procedure

Spontaneous intrahepatic portosystemic

venous shunt

Steatohepatitis

Stomal varices

Subacute hepatic failure

Sugiura procedure

Suspected drug-induced liver injury<sup>1</sup>

Transient hepatic attenuation differences

Varices oesophageal

Varicose veins of abdominal wall

White nipple sign

Liver function test abnormal

Liver function test decreased

Liver function test increased

Liver induration

Liver iron concentration abnormal

Liver iron concentration increased

Liver opacity



Hepatic cancer stage II Liver palpable

Hepatic cancer stage III Liver scan abnormal

Hepatic cancer stage IV Liver tenderness

Hepatic cirrhosis Magnetic resonance imaging hepatobiliary

abnormal

Hepatic cyst

Magnetic resonance proton density fat

fraction measurement

Hepatic cyst ruptured Mitochondrial aspartate aminotransferase

increased

Hepatic cytolysis

Model for end stage liver disease score

abnormal

Hepatic encephalopathy Model for end stage liver disease score

increased

Hepatic encephalopathy prophylaxis

Molar ratio of total branched-chain amino

acid to tyrosine

Hepatic failure Osteopontin increased

Hepatic fibrosis Perihepatic discomfort

Hepatic haemangioma rupture Periportal oedema

Hepatic hamartoma Peritoneal fluid protein abnormal

Hepatic hydrothorax Peritoneal fluid protein decreased

Hepatic infiltration eosinophilic Peritoneal fluid protein increased

Hepatic lesion Pneumobilia

Hepatic necrosis Portal vein flow decreased

Hepatic neoplasm Portal vein pressure increased

Hepatic perfusion disorder Retinol binding protein decreased

Hepatic steato-fibrosis Transaminases abnormal<sup>1</sup>

Hepatic steatosis Transaminases increased<sup>1</sup>

Hepatitis Ultrasound liver abnormal

Hepatitis acute Urine bilirubin increased



Hepatitis chronic active

Hepatitis chronic persistent

Hepatitis fulminant

Hepatitis toxic<sup>1</sup>

Guanase increased

Haemorrhagic ascites

Hepaplastin abnormal

Hepaplastin decreased

Hepatic artery flow decreased

Hepatic enzyme abnormal

Hepatic enzyme decreased

Hepatic enzyme increased

Hepatic fibrosis marker abnormal

Hepatic fibrosis marker increased

Hepatic function abnormal

Hepatic hypertrophy

<sup>1</sup>Narrow term.

Urobilinogen urine decreased

Urobilinogen urine increased

X-ray hepatobiliary abnormal

Protein C decreased

Protein S abnormal

Protein S decreased

Prothrombin level abnormal

Prothrombin level decreased

Prothrombin time abnormal

Prothrombin time prolonged

Prothrombin time ratio abnormal

Prothrombin time ratio increased

# 8.4.1.4. Electrolyte Disorder

Selected treatment-emergent abnormally low electrolyte disorder adverse events will be summarized. The electrolyte disorder search definition is a custom MedDRA version 27.0 query based on selected terms from the Metabolism and nutrition disorders and Investigations SOCs. The PTs are as defined below for each electrolyte. The frequency table will be summarized by descending frequency of lab analyte and PT. A shift table will be generated for lab grades in hypocalcemia, hypercalcemia, hypomagnesemia, hypermagnesemia, hypokalemia, hyperkalemia, hyponatremia, and hypernatremia, as well as for clinical categorization in phosphate.



**Lab Analyte Pertinent PTs** 

Hypocalcaemia: Blood calcium decreased, Hypocalcaemia, Hypocalcaemic seizure

Hypomagnesaemia: Blood magnesium decreased, Hypomagnesaemia

Hypophosphatemia: Blood phosphorus decreased, Hypophosphataemia

Hypokalaemia: Blood potassium decreased, Hypokalaemia, Hypokalaemic

syndrome

Blood sodium decreased, Hyponatraemia, Hyponatraemic coma,

Hyponatraemic encephalopathy, Hyponatraemic seizure,

Hyponatraemic syndrome

#### 8.4.1.5. Non-Melanoma Skin Cancers

The non-melanoma skin cancers search definition is a custom MedDRA version 27.0 query based on selected terms from the Skin neoplasms malignant and unspecified (excluding melanoma) HLT within the Neoplasms benign, malignant and unspecified (including cysts and polyps) SOC, plus the PT of Squamous cell carcinoma. The PTs are shown below:

Atypical fibroxanthoma Neoplasm skin

Basal cell carcinoma Neuroendocrine carcinoma of the skin

Basal cell carcinoma metastatic Pilomatrix carcinoma

Basal cell naevus syndrome Porocarcinoma

Basosquamous carcinoma of skin Primary cutaneous adenoid cystic carcinoma

Bowen's disease Sebaceous carcinoma

Carcinoma in situ of skin Squamoproliferative lesion

Dysplastic naevus syndrome Skin angiosarcoma

Eccrine carcinoma Skin cancer

Epidermal naevus syndrome Skin cancer metastatic

Keratoacanthoma Skin neoplasm bleeding

Malignant sweat gland neoplasm Skin squamous cell carcinoma metastatic



Marjolin's ulcer Skin squamous cell carcinoma recurrent

Mastocytoma Squamous cell carcinoma of skin

Trichoblastic carcinoma

Squamous cell carcinoma

# 8.4.2. Other Safety Topics of Special Interest

Safety topics of special interest have been identified based on the review of safety data from prior studies with nirogacestat and include additional AEs beyond those specified in Protocol Section 11.3.1 as AESIs. These safety topics of interest are defined for analysis purposes by using standardized MedDRA queries (SMQ) or customized MedDRA queries, as described below.

#### 8.4.2.1. Musculoskeletal Disorders

The Musculoskeletal Disorders search definition is a custom MedDRA version 27.0 query based on selected terms from the Bone disorders (excluding congenital and fractures) HLGT. The PTs are shown below:

Bone atrophy Fracture delayed union

Bone callus excessive Fracture malunion

Bone decalcification Fracture nonunion

Bone erosion Idiopathic juvenile osteoporosis

Bone demineralisation Melorheostosis

Bone formation decreased Osteodystrophy

Bone formation increased Osteolysis

Bone hypertrophy Osteomalacia

Bone loss Osteopenia

Bone pain Osteoporosis

Callus formation delayed Osteoporosis circumscripta cranii

Enostosis Osteoporosis postmenopausal



Exostosis Osteosclerosis

Exostosis of external ear canal Osteosis

Exostosis of jaw Resorption bone decreased

Extraskeletal ossification Resorption bone increased

#### 8.4.2.2. Bone Fracture

The Bone Fracture search definition is a custom MedDRA version 27.0 query based on selected terms from the Fractures of the Musculoskeletal HLGT and Connective tissue disorders SOC. The PTs are shown below:

Acetabulum fracture Impacted fracture

Ankle fracture Jaw fracture

Atypical femur fracture Limb fracture

Atypical fracture Lisfranc fracture

Avulsion fracture Lower limb fracture

Bone fissure Lumbar vertebral fracture

Bone fragmentation Maisonneuve fracture

Cervical vertebral fracture Metaphyseal corner fracture

Chance fracture Multiple fractures

Clavicle fracture Neurogenic fracture

Comminuted fracture Open fracture

Complicated fracture Osteochondral fracture

Compression fracture Osteo-meningeal breaches

Costal cartilage fracture Osteophyte fracture

Craniofacial fracture Osteoporotic fracture

Craniofacial injury Patella fracture

Epiphyseal fracture Pathological fracture

Facial bones fracture Pelvic fracture



Femoral neck fracture Periprosthetic fracture

Femur fracture Pseudarthrosis

Fibula fracture Pseudofracture

Flail chest Radius fracture

Foot fracture Rib fracture

Forearm fracture Sacroiliac fracture

Fracture Scapula fracture

Fracture blisters Scapulothoracic dissociation

Fracture delayed union Skull fracture

Fracture displacement Skull fractured base

Fracture infection Spinal compression fracture

Fracture malunion Spinal fracture

Fracture nonunion Spinal fusion fracture

Fracture of clavicle due to birth trauma

Sternal fracture

Fractured coccyx Stress fracture

Fractured sacrum Subchondral insufficiency fracture

Fractured skull depressed Thoracic vertebral fracture

Greenstick fracture Tibia fracture

Hand fracture Torus fracture

Hip fracture Traumatic fracture

Humerus fracture Ulna fracture

Ilium fracture Upper limb fracture

Wrist fracture



# 8.4.2.3. Mucositis/Stomatitis

The Mucositis/Stomatitis search definition is a custom MedDRA version 27.0 query based on selected terms from the Stomatitis and ulceration and Oral soft tissue signs and symptoms HLTs. The PTs are shown below:

Mouth ulceration Palatal ulcer

Oral mucosa erosion Stomatitis haemorrhagic

Oral pain Stomatitis necrotizing

Oropharyngeal pain Stomatitis

# 8.4.2.4. Hematologic Disorders

The Hematologic Disorders search definition is a custom MedDRA version 27.0 query based on selected terms from the Blood and lymphatic disorders SOC. The PTs are shown below:

Agranulocytosis Lymphocyte percentage decreased

Anaemia Lymphocytopenia neonatal

Anaemia macrocytic Lymphopenia

Anaemia neonatal Metamyelocyte count decreased

Aplasia pure red cell Microcytic anaemia

Aplastic anaemia Monoblast count decreased

Band neutrophil count decreased Monocyte count abnormal

Band neutrophil percentage decreased Monocyte count decreased

Basophil count abnormal Monocyte percentage decreased

Basophil count decreased Monocytopenia

Basophil percentage decreased Mononuclear cell count decreased

Basophilopenia Myeloblast count decreased

B-lymphocyte abnormalities Myeloblast percentage decreased

B-lymphocyte count abnormal Myelocyte count decreased

B-lymphocyte count decreased Myelocyte percentage decreased

Cyclic neutropenia Myeloid maturation arrest



Differential white blood cell count

abnormal

Neutropenia

Eosinopenia Neutropenia neonatal

Eosinophil count abnormal Neutropenic infection

Eosinophil count decreased Neutropenic sepsis

Eosinophil percentage decreased Neutrophil count abnormal

Erythroblast count abnormal Neutrophil count decreased

Erythroblast count decreased Neutrophil percentage decreased

Erythroid maturation arrest Normochromic anaemia

Erythropenia Normochromic normocytic anaemia

Erythropoiesis abnormal Normocytic anaemia

Febrile neutropenia Plasma cell disorder

Foetal anaemia Plasma cells absent

Full blood count abnormal Proerythroblast count abnormal

Granulocyte count decreased Proerythroblast count decreased

Granulocytes abnormal Promyelocyte count decreased

Granulocytes maturation arrest Pure white cell aplasia

Granulocytopenia Radiation leukopenia

Granulocytopenia neonatal Red blood cell count abnormal

Haematocrit abnormal Red blood cell count decreased

Haematocrit decreased Reticulocyte count abnormal

Haemoglobin abnormal Reticulocyte count decreased

Haemoglobin decreased Reticulocyte percentage decreased

Hypohaemoglobinaemia Reticulocytopenia

Hypoplastic anaemia T-lymphocyte count abnormal

Idiopathic neutropenia T-lymphocyte count abnormal

Leukoerythroblastic anaemia T-lymphocyte count decreased


Leukopenia White blood cell analysis abnormal

Leukopenia neonatal White blood cell count abnormal

Lymphocyte count abnormal White blood cell count decreased

Lymphocyte count decreased White blood cell disorder

Lymphocyte percentage abnormal

# 8.4.2.5. Opportunistic Infections

The Opportunistic Infections search definition is based on MedDRA version 27.0 Narrow and Broad terms from the Opportunistic Infections SMQ. The PTs are shown below, with Narrow search terms indicated:

Abdominal sepsis Human herpesvirus 6 infection reactivation<sup>1</sup>

Abiotrophia defectiva endocarditis<sup>1</sup> Human herpesvirus 6 viraemia<sup>1</sup>

Abscess fungal Human herpesvirus 7 infection

Acanthamoeba infection Human herpesvirus 8 infection<sup>1</sup>

Achromobacter infection Human metapneumovirus test positive

Acid fast bacilli infection<sup>1</sup> Human papilloma virus test positive

Acinetobacter bacteraemia Human polyomavirus infection

Hyperparasitaemia<sup>1</sup>

Acinetobacter infection Immune reconstitution inflammatory syndrome

Acinetobacter sepsis<sup>1</sup> Immune reconstitution inflammatory syndrome

associated tuberculosis<sup>1</sup>

Actinomyces test positive Indeterminate leprosy<sup>1</sup>

Indeterminate tuberculosis test

Actinomycosis Infection in an immunocompromised host<sup>1</sup>

Actinomycotic abdominal infection Infection susceptibility increased<sup>1</sup>

Actinomycotic pulmonary infection Infectious thyroiditis

Actinomycotic sepsis<sup>1</sup> Infective aneurysm



Actinomycotic skin infection Influenza

Acute haemorrhagic conjunctivitis Influenza A virus test positive

Acute hepatitis B Influenza B virus test positive

Acute hepatitis C Influenza C virus test positive

Influenza myocarditis

Acute pulmonary histoplasmosis<sup>1</sup> Influenza virus test positive

Adenoviral conjunctivitis Interferon gamma release assay positive

Adenoviral encephalitis<sup>1</sup> Intestinal tuberculosis<sup>1</sup>

Adenoviral haemorrhagic cystitis<sup>1</sup> Isosporiasis<sup>1</sup>

Jamestown Canyon encephalitis

Adenoviral hepatitis JC polyomavirus test positive

Adenoviral meningitis<sup>1</sup> JC virus CSF test positive<sup>1</sup>

Adenoviral upper respiratory infection JC virus granule cell neuronopathy<sup>1</sup>

Adenovirus

encephalomyeloradiculitis<sup>1</sup>

JC virus infection<sup>1</sup>

Adenovirus infection Joint tuberculosis<sup>1</sup>

Adenovirus interstitial nephritis<sup>1</sup>

Adenovirus test positive Kaposi's sarcoma<sup>1</sup>

Adrenal gland tuberculosis<sup>1</sup> Kaposi's sarcoma AIDS related<sup>1</sup>

Aerococcus urinae infection Keratitis fungal

Aeromonas infection Keratitis viral

Aeromonas test positive Klebsiella bacteraemia

African trypanosomiasis Klebsiella infection

Klebsiella pneumoniae invasive syndrome

Alcaligenes infection Klebsiella sepsis

Algid malaria

Allergic bronchopulmonary mycosis Klebsiella test positive



Lactobacillus bacteraemia

Allescheriosis Lactobacillus infection

Alpha haemolytic streptococcal

infection

Laryngeal cryptococcosis<sup>1</sup>

Alphavirus test positive Laryngitis fungal<sup>1</sup>

Leclercia bacteraemia<sup>1</sup>

Alternaria infection Legionella infection

American trypanosomiasis Legionella test positive

Amoeba test positive Leishmaniasis

Amoebiasis Lepromatous leprosy<sup>1</sup>

Amoebic brain abscess<sup>1</sup> Leprosy<sup>1</sup>

Amoebic colitis Leptotrichia infection

Amoebic dysentery Leuconostoc infection

Amoebic lung abscess<sup>1</sup> Listeria encephalitis<sup>1</sup>

Amoebic skin ulcer Listeria sepsis<sup>1</sup>

Amoeboma<sup>1</sup>

Anal candidiasis Listeria test positive

Anal fungal infection Listeriosis<sup>1</sup>

Angina gangrenous Lower respiratory tract herpes infection<sup>1</sup>

Angiostrongylus infection Lower respiratory tract infection fungal<sup>1</sup>

Anogenital warts Lower respiratory tract infection viral

Anorectal human papilloma virus

infection

Lupus vulgaris<sup>1</sup>

Anthrax sepsis Lymph node tuberculosis<sup>1</sup>

Anti-JC virus antibody index Lymphadenitis fungal<sup>1</sup>

Arbovirus test positive Malaria

Arenavirus test positive Malaria antibody test positive

Arthritis fungal<sup>1</sup> Malarial myocarditis



Arthritis salmonella Male genital tract tuberculosis<sup>1</sup>

Arthritis-dermatitis syndrome

Aspergilloma Mammary tuberculosis<sup>1</sup>

Aspergillosis oral<sup>1</sup> Mastitis fungal<sup>1</sup>

Mastoiditis fungal

Aspergillus infection<sup>1</sup> Measles meningitis

Aspergillus test positive Meningitis aspergillus<sup>1</sup>

Atypical mycobacterial infection<sup>1</sup> Meningitis candida<sup>1</sup>

Atypical mycobacterial lower respiratory tract infection<sup>1</sup> Meningitis coccidioides<sup>1</sup>

Atypical mycobacterial

lymphadenitis<sup>1</sup>

Meningitis cronobacter

Atypical mycobacterial pneumonia<sup>1</sup> Meningitis cryptococcal<sup>1</sup>

Atypical mycobacterium pericarditis<sup>1</sup> Meningitis enterococcal

Atypical mycobacterium test positive Meningitis exserohilum<sup>1</sup>

Atypical pneumonia Meningitis fungal<sup>1</sup>

Avian influenza Meningitis haemophilus

Babesiosis Meningitis herpes<sup>1</sup>

Bacillary angiomatosis<sup>1</sup> Meningitis histoplasma<sup>1</sup>

Bacteraemia Meningitis listeria<sup>1</sup>

Bacterial myositis Meningitis meningococcal

Bacterial sepsis Meningitis pneumococcal

Bacterial test positive Meningitis salmonella

Balamuthia infection Meningitis staphylococcal

Balanitis candida Meningitis streptococcal

Bartonella test positive Meningitis toxoplasmal<sup>1</sup>

Bartonellosis Meningitis trypanosomal



Beta haemolytic streptococcal

infection

Meningitis tuberculous<sup>1</sup>

Biliary sepsis Meningoencephalitis herpes simplex neonatal

Biliary tract infection cryptosporidial<sup>1</sup>

Biliary tract infection fungal<sup>1</sup> Meningoencephalitis viral

BK polyomavirus test positive Meningomyelitis herpes<sup>1</sup>

BK virus infection Merkel cell polyomavirus infection

Bladder candidiasis MERS-CoV test positive

Blastocystis infection<sup>1</sup> Metapneumovirus bronchiolitis

Blastomycosis<sup>1</sup> Metapneumovirus infection

Blood beta-D-glucan abnormal Metapneumovirus pneumonia

Blood beta-D-glucan increased Methylobacterium infection<sup>1</sup>

Blood beta-D-glucan positive Micrococcal sepsis

Blood culture positive Micrococcus infection

Body tinea Micrococcus test positive

Bone tuberculosis<sup>1</sup> Microsporidia infection<sup>1</sup>

Borderline leprosy<sup>1</sup> Microsporum infection

Botryomycosis Middle East respiratory syndrome

Bovine tuberculosis<sup>1</sup> Miliary pneumonia<sup>1</sup>

Breakthrough COVID-19

Bronchitis fungal<sup>1</sup> Morganella infection

Bronchitis haemophilus Mucocutaneous candidiasis

Bronchopulmonary aspergillosis<sup>1</sup> Mucormycosis<sup>1</sup>

Multisystem inflammatory syndrome in adults

Bronchopulmonary aspergillosis

allergic

Multisystem inflammatory syndrome in children

Brucella sepsis Mumps antibody test positive

Brucella test positive Murray Valley encephalitis



Bullous impetigo Mycetoma mycotic<sup>1</sup>

Burkholderia cepacia complex

infection

Mycobacterial infection<sup>1</sup>

Burkholderia cepacia complex sepsis<sup>1</sup> M

Mycobacterial peritonitis<sup>1</sup>

Burkholderia gladioli infection<sup>1</sup>

Mycobacterium abscessus infection<sup>1</sup>

Burkholderia infection

Mycobacterium avium complex immune restoration

disease<sup>1</sup>

Burkholderia mallei infection

Mycobacterium avium complex infection<sup>1</sup>

Burkholderia pseudomallei infection<sup>1</sup>

Mycobacterium chelonae infection<sup>1</sup>

Burkholderia test positive

Mycobacterium fortuitum infection<sup>1</sup>

Bursitis infective staphylococcal

Mycobacterium kansasii infection<sup>1</sup>

Buschke-Lowenstein's tumour

Mycobacterium leprae test positive

Cache Valley virus infection

Campylobacter bacteraemia

Campylobacter sepsis Mycobacterium marinum infection<sup>1</sup>

Campylobacter test positive

Mycobacterium test positive

Candida cervicitis

Mycobacterium tuberculosis complex test positive

Candida endophthalmitis<sup>1</sup>

Mycobacterium ulcerans infection<sup>1</sup>

Candida infection

Mycotic corneal ulcer

Candida osteomyelitis<sup>1</sup>

Mycotic endophthalmitis<sup>1</sup>

Candida pneumonia<sup>1</sup>

Mycotoxicosis

Candida retinitis<sup>1</sup>

Myocarditis mycotic<sup>1</sup>

Candida sepsis<sup>1</sup>

Myocarditis septic

Candida test positive

Myocarditis toxoplasmal<sup>1</sup>

Candidiasis of trachea<sup>1</sup>

Nail candida

Capnocytophaga infection<sup>1</sup>

Nasal candidiasis

Capnocytophaga sepsis<sup>1</sup>

Nasal herpes

Capnocytophaga test positive

Necrotising fasciitis fungal<sup>1</sup>



Capripox viral infection

Cardiac tuberculosis<sup>1</sup>

Cat scratch disease Necrotising fasciitis staphylococcal

Cellulitis enterococcal Necrotising fasciitis streptococcal

Cellulitis pasteurella Necrotising herpetic retinopathy<sup>1</sup>

Cellulitis staphylococcal Neisseria test positive

Neonatal bacteraemia

Cellulitis streptococcal Neonatal candida infection

Central nervous system fungal

infection<sup>1</sup>

Neonatal infective mastitis

Central nervous system listeria

infection<sup>1</sup>

Central nervous system viral

infection<sup>1</sup>

Neonatal mucocutaneous herpes simplex

Cerebral aspergillosis<sup>1</sup> Neurocryptococcosis<sup>1</sup>

Cerebral fungal infection<sup>1</sup> Neutropenic infection

Cerebral malaria Neutropenic sepsis<sup>1</sup>

Cerebral nocardiosis<sup>1</sup>

Cerebral toxoplasmosis<sup>1</sup> Nocardia sepsis<sup>1</sup>

Cervicitis human papilloma virus Nocardia test positive

Cervicitis streptococcal Nocardiosis<sup>1</sup>

Cervix warts Oesophageal candidiasis<sup>1</sup>

Chagas' cardiomyopathy

Chagas' gastrointestinal disease

Chancroid Oesophageal tuberculosis<sup>1</sup>

Chlamydia test positive Onychomycosis

Choriomeningitis lymphocytic Ophthalmic herpes simplex<sup>1</sup>

Choroid tubercles<sup>1</sup> Ophthalmic herpes zoster<sup>1</sup>



Chromoblastomycosis<sup>1</sup> Opportunistic infection<sup>1</sup>

Chronic active Epstein-Barr virus

infection

Oral candidiasis

Chronic hepatitis B Oral fungal infection

Chronic hepatitis C Oral hairy leukoplakia

Chronic hyperplastic candidiasis<sup>1</sup>

Chronic pulmonary histoplasmosis<sup>1</sup> Oral herpes

Oral herpes zoster

Citrobacter infection Oral tuberculosis<sup>1</sup>

Citrobacter sepsis Organic dust toxic syndrome

Citrobacter test positive Oro-pharyngeal aspergillosis<sup>1</sup>

Clostridial sepsis Oropharyngeal candidiasis

Clostridium bacteraemia Oropharyngitis fungal

Clostridium colitis Orthopox virus infection

Clostridium difficile colitis Orthopoxvirus test positive

Osteoarticular sporotrichosis<sup>1</sup>

Clostridium difficile infection Osteomyelitis blastomyces<sup>1</sup>

Clostridium test positive Osteomyelitis fungal<sup>1</sup>

Coccidioides encephalitis<sup>1</sup> Osteomyelitis salmonella

Coccidioidomycosis<sup>1</sup> Otitis externa candida

Colitis herpes<sup>1</sup> Otitis media fungal<sup>1</sup>

Complicated malaria

Conjunctivitis tuberculous<sup>1</sup> Otitis media haemophilus

Coronavirus infection

Coronavirus pneumonia

Coronavirus test positive Pancreatitis fungal<sup>1</sup>

Corynebacterium infection Pantoea agglomerans infection



Corynebacterium sepsis Pantoea agglomerans test positive

Corynebacterium test positive Papilloma viral infection

COVID-19 Paracoccidioides infection<sup>1</sup>

COVID-19 pneumonia Parainfluenzae viral bronchitis

Coxiella infection Parainfluenzae viral laryngotracheobronchitis

Coxiella test positive Parainfluenzae virus infection

Coxsackie viral disease of the

newborn

Parapharyngeal space infection

Creutzfeldt-Jakob disease Parasitic encephalitis

Cronobacter bacteraemia Parechovirus infection

Cronobacter infection Parvovirus B19 infection reactivation<sup>1</sup>

Cronobacter necrotising enterocolitis Pasteurella test positive

Cryptococcal cutaneous infection<sup>1</sup> Peliosis hepatis

Cryptococcal fungaemia<sup>1</sup> Pelvic sepsis

Cryptococcal meningoencephalitis<sup>1</sup> Penicillium infection<sup>1</sup>

Cryptococcosis<sup>1</sup> Penile gangrene

Cryptococcus test positive Penile wart

Cryptosporidiosis infection Peptostreptococcus infection

CSF measles antibody positive Peptostreptococcus test positive

Cutaneous anthrax Perianal streptococcal infection

Cutaneous coccidioidomycosis<sup>1</sup> Pericarditis fungal<sup>1</sup>

Cutaneous mucormycosis Pericarditis histoplasma<sup>1</sup>

Cutaneous sporotrichosis Pericarditis tuberculous<sup>1</sup>

Cutaneous tuberculosis<sup>1</sup> Perinatal HBV infection

Cyclosporidium infection Periporitis staphylogenes

Cystitis escherichia Peritoneal candidiasis<sup>1</sup>

Cystitis klebsiella Peritoneal tuberculosis<sup>1</sup>



Cystitis pseudomonal Peritonitis pneumococcal

Cytomegalovirus chorioretinitis<sup>1</sup> Phaeohyphomycosis<sup>1</sup>

Cytomegalovirus colitis<sup>1</sup> Pharyngeal abscess

Cytomegalovirus duodenitis<sup>1</sup> Pharyngoconjunctival fever of children

Cytomegalovirus enteritis<sup>1</sup> Plasmodium falciparum infection

Cytomegalovirus enterocolitis<sup>1</sup> Plasmodium malariae infection

Cytomegalovirus gastritis<sup>1</sup> Plasmodium ovale infection

Cytomegalovirus gastroenteritis<sup>1</sup> Plasmodium vivax infection

Plesiomonas shigelloides infection

Cytomegalovirus gastrointestinal

infection<sup>1</sup>

Pneumococcal bacteraemia

Cytomegalovirus gastrointestinal

ulcerl

Pneumococcal infection

Cytomegalovirus hepatitis<sup>1</sup> Pneumococcal sepsis

Cytomegalovirus immunisation Pneumocystis jirovecii infection<sup>1</sup>

Cytomegalovirus infection<sup>1</sup> Pneumocystis jirovecii pneumonia<sup>1</sup>

Cytomegalovirus infection

reactivation<sup>1</sup>

Pneumocystis test positive

Cytomegalovirus mononucleosis<sup>1</sup> Pneumonia adenoviral

Cytomegalovirus mucocutaneous

ulcer1

Pneumonia anthrax

Cytomegalovirus

myelomeningoradiculitis<sup>1</sup>

Cytomegalovirus myocarditis<sup>1</sup> Pneumonia cryptococcal<sup>1</sup>

Cytomegalovirus oesophagitis<sup>1</sup> Pneumonia cytomegaloviral<sup>1</sup>

Cytomegalovirus pancreatitis<sup>1</sup> Pneumonia escherichia

Cytomegalovirus pericarditis<sup>1</sup> Pneumonia fungal<sup>1</sup>

Cytomegalovirus syndrome<sup>1</sup> Pneumonia haemophilus

Cytomegalovirus test positive Pneumonia herpes viral<sup>1</sup>



Cytomegalovirus urinary tract

infection<sup>1</sup>

Pneumonia influenzal

Cytomegalovirus viraemia<sup>1</sup>

Pneumonia Klebsiella

Delftia acidovorans infection

Pneumonia legionella<sup>1</sup>

Deltaretrovirus test positive

Pneumonia measles

Dengue fever

Pneumonia parainfluenzae viral

Dengue shock syndrome

Dental sepsis

Dermatolymphangioadenitis

Device related bacteraemia

Pneumonia pneumococcal

Device related fungaemia

Device related sepsis

Pneumonia pseudomonal

Disseminated aspergillosis<sup>1</sup>

Pneumonia respiratory syncytial viral

Disseminated blastomycosis<sup>1</sup>

Pneumonia salmonella

Disseminated coccidioidomycosis<sup>1</sup>

Pneumonia staphylococcal

Disseminated cryptococcosis<sup>1</sup>

Pneumonia streptococcal

Disseminated cytomegaloviral

infection<sup>1</sup>

Pneumonia toxoplasmal<sup>1</sup>

Disseminated enteroviral infection<sup>1</sup>

Disseminated gonococcal infection

Disseminated herpes simplex

Disseminated leishmaniasis<sup>1</sup>

Polyomavirus test positive

Disseminated mucormycosis<sup>1</sup>

Polyomavirus viraemia<sup>1</sup>

Disseminated mycobacterium avium

complex infection<sup>1</sup>

Polyomavirus-associated nephropathy1

Disseminated

paracoccidioidomycosis<sup>1</sup>

Pontiac fever

Porphyromonas bacteraemia



Disseminated sporotrichosis<sup>1</sup> Porphyromonas infection

Disseminated strongyloidiasis<sup>1</sup> Porphyromonas test positive

Disseminated toxoplasmosis<sup>1</sup> Post streptococcal glomerulonephritis

Disseminated trichosporonosis<sup>1</sup> Post transplant lymphoproliferative disorder

Disseminated tuberculosis<sup>1</sup> Presumed ocular histoplasmosis syndrome

Disseminated varicella<sup>1</sup> Prion agent test positive

Disseminated varicella zoster vaccine

virus infection<sup>1</sup>

Proctitis fungal

Disseminated varicella zoster virus

infection1

Proctitis herpes<sup>1</sup>

Ear infection fungal Proctitis monilial

Ear tuberculosis<sup>1</sup> Progressive multifocal leukoencephalopathy<sup>1</sup>

Eczema herpeticum Progressive vaccinia<sup>1</sup>

Elsberg syndrome<sup>1</sup>

Encephalitis australia Prostatitis Escherichia coli

Encephalitis california Prostatitis tuberculous<sup>1</sup>

Encephalitis cytomegalovirus<sup>1</sup> Protothecosis<sup>1</sup>

Encephalitis eastern equine Pseudallescheria infection<sup>1</sup>

Encephalitis enteroviral Pseudallescheria sepsis<sup>1</sup>

Encephalitis fungal<sup>1</sup> Pseudoaneurysm infection

Encephalitis herpes<sup>1</sup>

Encephalitis influenzal Pseudomonal bacteraemia

Encephalitis Japanese B Pseudomonal sepsis

Encephalitis meningococcal Pseudomonas aeruginosa meningitis<sup>1</sup>

Encephalitis mumps Pseudomonas bronchitis

Encephalitis post varicella<sup>1</sup> Pseudomonas infection

Encephalitis protozoal Pseudomonas peritonitis

Encephalitis rickettsial Pseudomonas test positive



Pulmonary blastomycosis<sup>1</sup>

Pulmonary gangrene

Pulmonary histoplasmosis<sup>1</sup>

Encephalitis venezuelan equine Pulmonary mucormycosis<sup>1</sup>

Encephalitis viral Pulmonary nocardiosis<sup>1</sup>

Encephalitis western equine Pulmonary sepsis

Encephalomyelitis rubella Pulmonary trichosporonosis<sup>1</sup>

Endocarditis candida<sup>1</sup> Pulmonary tuberculoma<sup>1</sup>

Endocarditis enterococcal Pulmonary tuberculosis<sup>1</sup>

Endocarditis haemophilus Pyelonephritis fungal<sup>1</sup>

Endocarditis histoplasma<sup>1</sup> Pyoderma streptococcal

Endocarditis pseudomonal Pythium insidiosum infection

Endocarditis Q fever<sup>1</sup> Q fever

Endocarditis staphylococcal Raoultella ornithinolytica infection

Endocarditis viral Renal tuberculosis<sup>1</sup>

Enterobacter bacteraemia Respiratory moniliasis

Enterobacter infection Respiratory syncytial virus bronchiolitis

Enterobacter pneumonia Respiratory syncytial virus bronchitis

Enterobacter sepsis Respiratory syncytial virus infection

Enterobacter test positive Respiratory syncytial virus test positive

Enterobacter tracheobronchitis Respiratory tract infection fungal<sup>1</sup>

Enterococcal bacteraemia Retinitis histoplasma<sup>1</sup>

Enterococcal infection Retinitis viral<sup>1</sup>

Enterococcal sepsis Retroviral rebound syndrome

Enterococcus test positive Rhinocerebral mucormycosis<sup>1</sup>

Rhizobium radiobacter bacteraemia<sup>1</sup>

Enterocolitis fungal<sup>1</sup> Rhodococcus infection<sup>1</sup>



Enterocolitis viral Rhodococcus test positive

Enterovirus test positive Roseolovirus test positive

Epididymitis blastomyces<sup>1</sup> Rubella antibody positive

Epididymitis tuberculous<sup>1</sup> Salmonella bacteraemia

Epiglottitis haemophilus Salmonella sepsis

Epstein-Barr viraemia Salmonella test positive

Epstein-Barr virus antibody positive Salmonellosis

Epstein-Barr virus antigen positive Salpingitis tuberculous<sup>1</sup>

Epstein-Barr virus associated

lymphoma

SARS-CoV-1 test positive

Epstein-Barr virus associated lymphoproliferative disorder<sup>1</sup>

SARS-CoV-2 antibody test positive

Epstein-Barr virus infection SARS-CoV-2 sepsis

Epstein-Barr virus infection

reactivation1

SARS-CoV-2 test false negative

Epstein-Barr virus test positive SARS-CoV-2 test positive

Erysipelas Scarlet fever

Erythema induratum Scedosporium infection<sup>1</sup>

Escherichia bacteraemia Sepsis

Escherichia infection Sepsis neonatal

Escherichia sepsis Sepsis pasteurella

Escherichia test positive Sepsis syndrome

Escherichia urinary tract infection Septic arthritis haemophilus

Escherichia vaginitis Septic arthritis staphylococcal<sup>1</sup>

Exanthema subitum Septic arthritis streptobacillus

Exserohilum infection<sup>1</sup> Septic arthritis streptococcal

Septic cardiomyopathy

Septic cerebral embolism



Exserohilum test positive Septic coagulopathy

Extrapulmonary tuberculosis<sup>1</sup> Septic embolus

Septic endocarditis

Eye infection fungal Septic necrosis

Eye infection staphylococcal Septic phlebitis

Eye infection toxoplasmal<sup>1</sup> Septic pulmonary embolism

Eye infection viral Septic shock

Female genital tract tuberculosis<sup>1</sup> Serratia bacteraemia

Flavivirus test positive Serratia infection

Flavobacterium infection<sup>1</sup> Serratia sepsis

Flavobacterium test positive Serratia test positive

Fournier's gangrene<sup>1</sup> Severe acute respiratory syndrome

Fungaemia<sup>1</sup> Severe invasive streptococcal infection

Fungal abscess central nervous

system<sup>1</sup>

Shewanella algae bacteraemia

Fungal cystitis Shigella infection

Fungal endocarditis<sup>1</sup> Shigella test positive

Fungal infection Silicotuberculosis

Fungal labyrinthitis<sup>1</sup> Sinusitis aspergillus<sup>1</sup>

Fungal myositis<sup>1</sup>

Fungal oesophagitis<sup>1</sup> Sinusitis fungal<sup>1</sup>

Fungal paronychia Skin candida

Fungal peritonitis<sup>1</sup> Sphingomonas paucimobilis bacteraemia<sup>1</sup>

Fungal retinitis<sup>1</sup> Sphingomonas paucimobilis infection<sup>1</sup>

Fungal rhinitis<sup>1</sup> Spleen tuberculosis<sup>1</sup>

Fungal sepsis<sup>1</sup> Splenic candidiasis<sup>1</sup>

Fungal test positive Splenic infection fungal<sup>1</sup>



Fungal tracheitis<sup>1</sup> Sporotrichosis

Fusarium endocarditis<sup>1</sup>

Fusarium infection<sup>1</sup> Spotted fever rickettsia test positive

Gastric ulcer helicobacter St. Louis encephalitis

Gastritis fungal<sup>1</sup> Staphylococcal abscess

Gastritis herpes<sup>1</sup> Staphylococcal bacteraemia

Gastroenteritis adenovirus Staphylococcal impetigo

Gastroenteritis aeromonas Staphylococcal infection

Gastroenteritis cryptococcal<sup>1</sup> Staphylococcal mediastinitis

Gastroenteritis cryptosporidial<sup>1</sup> Staphylococcal osteomyelitis

Gastroenteritis Escherichia coli Staphylococcal scalded skin syndrome

Gastroenteritis pseudomonas Staphylococcal sepsis

Gastroenteritis salmonella Staphylococcal skin infection

Gastroenteritis staphylococcal Staphylococcal toxaemia

Gastroenteritis vibrio Staphylococcus test positive

Gastrointestinal anthrax Stenotrophomonas bacteraemia<sup>1</sup>

Gastrointestinal candidiasis Stenotrophomonas infection<sup>1</sup>

Stenotrophomonas maltophilia pneumonia<sup>1</sup>

Gastrointestinal fungal infection<sup>1</sup> Stenotrophomonas sepsis<sup>1</sup>

Gastrointestinal mucormycosis<sup>1</sup> Stenotrophomonas test positive

Genital candidiasis Stoma site candida

Genital herpes Stomatococcal infection

Genital herpes simplex Stomatococcus test positive

Genital herpes zoster Streptobacillary fever

Genital infection fungal Streptobacillus infection

Geotrichum infection Streptobacillus test positive

Group B streptococcus neonatal sepsis Streptococcal abscess



H1N1 influenza Streptococcal bacteraemia

Haematological infection

Haemophilus bacteraemia Streptococcal bronchitis

Haemophilus infection Streptococcal endocarditis

Haemophilus sepsis Streptococcal impetigo

Haemophilus test positive Streptococcal infection

Helicobacter gastritis Streptococcal sepsis

Helicobacter infection Streptococcal urinary tract infection

Helicobacter sepsis Streptococcus test positive

Helicobacter test positive Streptokinase antibody increased

Hepatic actinomycosis<sup>1</sup>

Hepatic candidiasis<sup>1</sup> Strongyloidiasis

Hepatic infection fungal<sup>1</sup> Subacute sclerosing panencephalitis

Submandibular abscess

Hepatitis A antibody abnormal Superinfection fungal<sup>1</sup>

Hepatitis A antibody positive Superinfection mycobacterial<sup>1</sup>

Hepatitis A antigen positive Suspected COVID-19

Hepatitis A virus test positive Syphilis

Syphilitic pelvic inflammatory disease<sup>1</sup>

Hepatitis B Systemic candida<sup>1</sup>

Hepatitis B antibody abnormal Systemic inflammatory response syndrome

Hepatitis B antibody positive Systemic mycosis<sup>1</sup>

Hepatitis B antigen positive Thrombophlebitis septic

Hepatitis B core antibody positive Thyroid tuberculosis<sup>1</sup>

Hepatitis B core antigen positive Tick-borne viral encephalitis

Hepatitis B DNA assay positive Tonsillitis fungal<sup>1</sup>

Hepatitis B DNA increased Torulopsis infection



Hepatitis B e antibody positive Toxic shock syndrome staphylococcal

Hepatitis B e antigen positive Toxic shock syndrome streptococcal

Hepatitis B surface antibody positive Toxoplasma serology positive

Hepatitis B surface antigen positive Toxoplasmosis<sup>1</sup>

Hepatitis B virus test positive Toxoplasmosis prophylaxis

Hepatitis C Treponema test positive

Hepatitis C antibody positive Trichophytic granuloma

Hepatitis C core antibody positive Trichosporon infection

Hepatitis C RNA increased Trypanosoma serology positive

Hepatitis C RNA positive Trypanosomiasis

Hepatitis C virus test positive Tuberculid

Hepatitis D Tuberculin test false negative

Hepatitis D antibody positive Tuberculin test false positive

Hepatitis D antigen positive Tuberculin test positive

Hepatitis D RNA positive Tuberculoid leprosy<sup>1</sup>

Tuberculoma<sup>1</sup>

Hepatitis D virus test positive Tuberculoma of central nervous system<sup>1</sup>

Hepatitis E antibody positive Tuberculosis<sup>1</sup>

Hepatitis E antigen positive Tuberculosis bladder<sup>1</sup>

Hepatitis E virus test positive Tuberculosis gastrointestinal<sup>1</sup>

Hepatitis infectious mononucleosis Tuberculosis liver<sup>1</sup>

Hepatitis non-A non-B Tuberculosis of central nervous system<sup>1</sup>

Hepatitis non-A non-B non-C Tuberculosis of eye<sup>1</sup>

Hepatitis syphilitic Tuberculosis of genitourinary system<sup>1</sup>

Hepatitis toxoplasmal Tuberculosis of intrathoracic lymph nodes<sup>1</sup>

Hepatitis viral test positive Tuberculosis of peripheral lymph nodes<sup>1</sup>

Tuberculosis of uterine cervix<sup>1</sup>



Hepatosplenic candidiasis<sup>1</sup> Tuberculosis ureter<sup>1</sup>

Herpes dermatitis Tuberculous abscess central nervous system<sup>1</sup>

Herpes gestationis Tuberculous endometritis<sup>1</sup>

Herpes oesophagitis<sup>1</sup> Tuberculous laryngitis<sup>1</sup>

Tuberculous pelvic inflammatory disease<sup>1</sup>

Herpes ophthalmic<sup>1</sup> Tuberculous pleurisy<sup>1</sup>

Herpes pharyngitis Tuberculous tenosynovitis<sup>1</sup>

Herpes sepsis<sup>1</sup> Typhus rickettsia test positive

Herpes simplex Upper respiratory fungal infection<sup>1</sup>

Herpes simplex bronchitis<sup>1</sup> Urinary tract candidiasis

Herpes simplex colitis<sup>1</sup> Urinary tract infection enterococcal

Herpes simplex encephalitis<sup>1</sup> Urinary tract infection fungal

Herpes simplex gastritis<sup>1</sup> Urinary tract infection pseudomonal

Herpes simplex hepatitis<sup>1</sup> Urinary tract infection staphylococcal

Herpes simplex meningitis<sup>1</sup> Urogenital infection fungal

Herpes simplex meningoencephalitis<sup>1</sup> Urosepsis

Herpes simplex meningomyelitis<sup>1</sup> Variant Creutzfeldt-Jakob disease

Herpes simplex necrotising

retinopathy1

Varicella

Varicella encephalitis<sup>1</sup>

Varicella meningitis<sup>1</sup>

Herpes simplex oesophagitis<sup>1</sup> Varicella post vaccine

Herpes simplex otitis externa<sup>1</sup> Varicella virus test positive

Herpes simplex pharyngitis Varicella zoster gastritis<sup>1</sup>

Herpes simplex pneumonia<sup>1</sup> Varicella zoster oesophagitis<sup>1</sup>

Herpes simplex sepsis<sup>1</sup> Varicella zoster pneumonia<sup>1</sup>

Herpes simplex test positive Varicella zoster sepsis<sup>1</sup>



Herpes simplex viraemia<sup>1</sup> Varicella zoster virus infection

Vascular access device culture positive

Herpes simplex virus conjunctivitis

neonatal

Vibrio test positive

Herpes simplex visceral<sup>1</sup> Viraemia

Herpes virus infection Viral myelitis

Herpes zoster Viral myocarditis

Herpes zoster cutaneous

disseminated1

Viral oesophagitis

Herpes zoster disseminated<sup>1</sup>

Herpes zoster infection neurological<sup>1</sup> Viral pericarditis

Herpes zoster meningitis<sup>1</sup> Viral sepsis

Herpes zoster meningoencephalitis<sup>1</sup> Viral test positive

Herpes zoster meningomyelitis<sup>1</sup> Viral uveitis

Herpes zoster meningoradiculitis<sup>1</sup> Visceral leishmaniasis<sup>1</sup>

Herpes zoster necrotising retinopathy<sup>1</sup> Vulvovaginal candidiasis

Herpes zoster oticus<sup>1</sup> Vulvovaginal human papilloma virus infection

Herpes zoster pharyngitis<sup>1</sup> Weissella infection<sup>1</sup>

Herpes zoster reactivation<sup>1</sup>

Histoplasmosis<sup>1</sup> West Nile viral infection

Histoplasmosis cutaneous<sup>1</sup> West Nile virus test positive

Histoplasmosis disseminated<sup>1</sup> Wound infection fungal

Human anaplasmosis Wound infection pseudomonas

Human ehrlichiosis Wound infection staphylococcal

Human herpes virus 6 serology

positive

Wound sepsis

WU virus infection

Human herpes virus 8 test positive Yersinia sepsis



Human herpesvirus 6 encephalitis<sup>1</sup>

Yersinia test positive

Zygomatic abscess

Human herpesvirus 6 infection

<sup>1</sup>Narrow term

## 8.4.2.6. Central Nervous System Vascular Disorders

The Central nervous system vascular disorders search definition is based on the MedDRA version 27.0 Narrow and Broad Terms from the Haemorrhagic central nervous system vascular conditions SMQ, Ischaemic central nervous system vascular conditions SMQ, and Central nervous system vascular disorders, not specified as haemorrhagic or ischaemic SMQ. The PTs are shown below, with Narrow search terms indicated:

Amaurosis fugax<sup>1</sup>

Amyloid related imaging abnormalities

Amyloid related imaging abnormality-microhaemorrhages

and haemosiderin deposits

Amyloid related imaging abnormality-oedema/effusion

Basal ganglia haematoma<sup>1</sup>

Basal ganglia haemorrhage<sup>1</sup>

Basal ganglia infarction<sup>1</sup>

Basal ganglia stroke1

Basilar artery occlusion<sup>1</sup>

Basilar artery perforation<sup>1</sup>

Basilar artery stenosis<sup>1</sup>

Basilar artery thrombosis<sup>1</sup>

Benedikt's syndrome<sup>1</sup>

Blood brain barrier defect

Brachiocephalic arteriosclerosis<sup>1</sup>

Brachiocephalic artery occlusion<sup>1</sup>

Brachiocephalic artery stenosis<sup>1</sup>

Brain hypoxia<sup>1</sup>

Brain stem embolism<sup>1</sup>

Cerebrovascular disorder<sup>1</sup> Cerebrovascular insufficiency<sup>1</sup>

Cerebrovascular stenosis<sup>1</sup>

Chronic cerebrospinal venous

insufficiency<sup>1</sup>

Claude's syndrome<sup>1</sup>

Congenital cerebrovascular

anomaly

Cortical hand stroke<sup>1</sup>

Delayed ischaemic neurological

deficit1

Dural arteriovenous fistula<sup>1</sup>

Embolic cerebellar infarction<sup>1</sup>

Embolic cerebral infarction<sup>1</sup>

Embolic stroke<sup>1</sup>

Extra-axial haemorrhage<sup>1</sup>
Extradural haematoma<sup>1</sup>
Extradural haematoma

evacuation<sup>1</sup>

Extraischaemic cerebral

haematoma1

Foetal cerebrovascular disorder<sup>1</sup>

Foville syndrome<sup>1</sup>

Haemorrhage intracranial<sup>1</sup>



Brain stem haematoma<sup>1</sup>

Brain stem haemorrhage<sup>1</sup>

Brain stem infarction<sup>1</sup>

Brain stem ischaemia<sup>1</sup>

Brain stem microhaemorrhage<sup>1</sup>

Brain stem stroke<sup>1</sup>

Brain stem thrombosis<sup>1</sup>

Brain stent insertion<sup>1</sup>

CADASIL<sup>1</sup>

Capsular warning syndrome<sup>1</sup>

CARASIL syndrome<sup>1</sup>

Carotid aneurysm rupture<sup>1</sup>

Carotid angioplasty<sup>1</sup>

Carotid arterial embolus<sup>1</sup>

Carotid arteriosclerosis<sup>1</sup>

Carotid artery bypass<sup>1</sup>

Carotid artery disease<sup>1</sup>

Carotid artery dolichoectasia

Carotid artery insufficiency<sup>1</sup>

Carotid artery occlusion<sup>1</sup>

Carotid artery perforation<sup>1</sup>

Carotid artery restenosis<sup>1</sup>

Carotid artery stenosis<sup>1</sup>

Carotid artery stent insertion<sup>1</sup>

Haemorrhagic cerebellar

infarction<sup>1</sup>

Haemorrhagic cerebral

infarction<sup>1</sup>

Haemorrhagic stroke<sup>1</sup>

Haemorrhagic transformation

stroke<sup>1</sup>

Hypertensive cerebrovascular

disease

Hypoxic-ischaemic encephalopathy<sup>1</sup>

Inner ear infarction<sup>1</sup>

Internal capsule infarction<sup>1</sup>

Intracerebral haematoma

evacuation1

Intracranial haematoma<sup>1</sup> Intracranial haemorrhage

neonatal1

Intracranial tumour

haemorrhage<sup>1</sup>

Intraventricular haemorrhage<sup>1</sup>

Intraventricular haemorrhage

neonatal1

Ischaemic cerebral infarction<sup>1</sup>

Ischaemic stroke<sup>1</sup>

Jugular vein embolism<sup>1</sup>

Lacunar infarction<sup>1</sup>

Lacunar stroke<sup>1</sup>

Lateral medullary syndrome<sup>1</sup>

Medullary compression

syndrome

Meningorrhagia<sup>1</sup>

Middle cerebral artery stroke<sup>1</sup>

Migrainous infarction<sup>1</sup>

Millard-Gubler syndrome<sup>1</sup>

Moyamoya disease<sup>1</sup>

Occipital lobe stroke<sup>1</sup>

Parietal lobe stroke<sup>1</sup>

Perinatal stroke<sup>1</sup>

Periventricular haemorrhage

neonatal<sup>1</sup>

Pituitary apoplexy<sup>1</sup>



Carotid artery stent removal<sup>1</sup> Carotid artery thrombosis<sup>1</sup> Carotid endarterectomy<sup>1</sup> Carotid revascularisation<sup>1</sup>

Central nervous system haemorrhage<sup>1</sup> Central nervous system vasculitis<sup>1</sup>

Cerebellar artery occlusion<sup>1</sup>

Cerebellar artery thrombosis<sup>1</sup>

Cerebellar atherosclerosis<sup>1</sup>

Cerebellar embolism<sup>1</sup>

Cerebellar haematoma<sup>1</sup>

Cerebellar haemorrhage<sup>1</sup>

Cerebellar infarction<sup>1</sup> Cerebellar ischaemia<sup>1</sup>

Cerebellar microhaemorrhage<sup>1</sup>

Cerebellar stroke1

Cerebral amyloid angiopathy

Cerebral aneurysm perforation<sup>1</sup>

Cerebral aneurysm ruptured syphilitic<sup>1</sup>

Cerebral angioplasty<sup>1</sup> Cerebral arteriosclerosis<sup>1</sup>

Cerebral arteriovenous malformation haemorrhagic<sup>1</sup>

Cerebral arteritis<sup>1</sup>

Cerebral artery embolism<sup>1</sup>

Cerebral artery occlusion<sup>1</sup> Cerebral artery perforation<sup>1</sup> Cerebral artery restenosis<sup>1</sup>

Cerebral artery stenosis<sup>1</sup>

Cerebral artery stent insertion<sup>1</sup> Cerebral artery thrombosis<sup>1</sup> Cerebral bypass surgery<sup>1</sup>

Pituitary haemorrhage<sup>1</sup>

Post cardiac arrest syndrome<sup>1</sup>

Post procedural stroke1

Precerebral arteriosclerosis<sup>1</sup>

Precerebral artery embolism<sup>1</sup>

Precerebral artery occlusion<sup>1</sup>

Precerebral artery thrombosis<sup>1</sup>

Primary familial brain

calcification

Pseudo-occlusion of internal

carotid artery<sup>1</sup>

Putamen haemorrhage<sup>1</sup>

Retinal artery occlusion<sup>1</sup>

Reversible cerebral

vasoconstriction syndrome<sup>1</sup>

Reversible ischaemic neurological deficit1

Ruptured cerebral aneurysm<sup>1</sup>

Sigmoid sinus thrombosis<sup>1</sup>

Sneddon's syndrome

Spinal artery embolism<sup>1</sup>

Spinal artery thrombosis<sup>1</sup>

Spinal cord haematoma<sup>1</sup>

Spinal cord haemorrhage<sup>1</sup>

Spinal cord hypoxia<sup>1</sup>

Spinal cord infarction<sup>1</sup>

Spinal cord ischaemia<sup>1</sup>

Spinal epidural haematoma<sup>1</sup>

Spinal epidural haemorrhage<sup>1</sup>

Spinal stroke<sup>1</sup>

Spinal subarachnoid

haemorrhage<sup>1</sup>

Spinal subdural haematoma<sup>1</sup>

Spinal subdural haemorrhage<sup>1</sup>

Spinal vascular disorder

Spinal vessel congenital

anomaly

Stroke in evolution<sup>1</sup>

Subarachnoid haematoma<sup>1</sup>



Cerebral capillary telangiectasia<sup>1</sup>

Cerebral circulatory failure<sup>1</sup>

Cerebral congestion<sup>1</sup>

Cerebral cyst haemorrhage<sup>1</sup>

Cerebral gas embolism<sup>1</sup>

Cerebral haematoma<sup>1</sup> Cerebral haemorrhage<sup>1</sup>

Cerebral haemorrhage foetal<sup>1</sup>

Cerebral haemorrhage neonatal<sup>1</sup>

Cerebral hypoperfusion<sup>1</sup>

Cerebral infarction<sup>1</sup>

Cerebral infarction foetal<sup>1</sup>

Cerebral ischaemia<sup>1</sup>

Cerebral microangiopathy Cerebral microembolism<sup>1</sup> Cerebral microhaemorrhage<sup>1</sup> Cerebral microinfarction<sup>1</sup> Cerebral revascularisation<sup>1</sup> Cerebral septic infarct<sup>1</sup>

Cerebral small vessel ischaemic disease<sup>1</sup>

Cerebral thrombosis<sup>1</sup>

Cerebral vascular occlusion<sup>1</sup>
Cerebral vasoconstriction<sup>1</sup>

Cerebral venous sinus thrombosis<sup>1</sup>

Cerebral venous thrombosis<sup>1</sup> Cerebrovascular accident<sup>1</sup>

Cerebrovascular arteriovenous malformation

<sup>1</sup>Narrow term.

Subarachnoid haemorrhage Subarachnoid haemorrhage

neonatal1

Subclavian steal syndrome<sup>1</sup>

Subcortical stroke<sup>1</sup>
Subdural haematoma<sup>1</sup>
Subdural haematoma

evacuation1

Subdural haemorrhage<sup>1</sup>

Subdural haemorrhage neonatal<sup>1</sup>

Superior sagittal sinus

thrombosis1

Susac's syndrome

Temporal artery stenosis<sup>1</sup>

Thalamic infarction<sup>1</sup>
Thalamic stroke<sup>1</sup>

Thalamus haemorrhage<sup>1</sup>

Thrombotic cerebral infarction<sup>1</sup>

Thrombotic stroke<sup>1</sup>

Transient ischaemic attack<sup>1</sup>
Transverse sinus thrombosis<sup>1</sup>
Vascular encephalopathy<sup>1</sup>
Vascular stent occlusion<sup>1</sup>
Vascular stent stenosis<sup>1</sup>

Vertebral artery arteriosclerosis<sup>1</sup>

Vertebral artery occlusion<sup>1</sup>
Vertebral artery perforation<sup>1</sup>
Vertebral artery stenosis<sup>1</sup>
Vertebral artery thrombosis<sup>1</sup>
Vertebrobasilar dolichoectasia
Vertebrobasilar infarction<sup>1</sup>
Vertebrobasilar insufficiency<sup>1</sup>

Vertebrobasilar stroke<sup>1</sup> Weber's syndrome<sup>1</sup>

#### 8.4.2.7. Embolic and Thrombotic Events

The Embolic and thrombotic events search definition is based on the MedDRA version 27.0 Embolic and thrombotic events, venous SMQ. The PTs are listed below, and all will be considered Narrow search terms:



Aseptic cavernous sinus thrombosis

Axillary vein thrombosis

Brachiocephalic vein occlusion

Brachiocephalic vein thrombosis

Budd-Chiari syndrome

Catheterisation venous

Cavernous sinus thrombosis

Central venous catheterisation

Cerebral venous sinus thrombosis

Cerebral venous thrombosis

Compression garment application

Deep vein thrombosis

Deep vein thrombosis postoperative

Embolism venous

Hepatic vein embolism

Hepatic vein occlusion

Hepatic vein thrombosis

Homans' sign positive

Iliac vein occlusion

Inferior vena cava syndrome

Inferior vena caval occlusion

Jugular vein embolism

Jugular vein occlusion

Jugular vein thrombosis

Mahler sign

May-Thurner syndrome

Mesenteric vein embolism

Mesenteric vein thrombosis

Mesenteric venous occlusion

Obstetrical pulmonary embolism

Obstructive shock

Ophthalmic vein thrombosis

Ovarian vein thrombosis

Pulmonary embolism

Pulmonary infarction

Pulmonary microemboli

Pulmonary oil microembolism

Pulmonary thrombosis

Pulmonary vein occlusion

Pulmonary veno-occlusive disease

Pulmonary venous thrombosis

Renal vein embolism

Renal vein occlusion

Renal vein thrombosis

Retinal vein occlusion

Retinal vein thrombosis

Septic pulmonary embolism

SI QIII TIII pattern

Sigmoid sinus thrombosis

Spermatic vein thrombosis

Splenic vein occlusion

Splenic vein thrombosis

Subclavian vein embolism

Subclavian vein occlusion

Subclavian vein thrombosis

Superior sagittal sinus thrombosis

Superior vena cava occlusion

Superior vena cava syndrome

Thrombophlebitis

Thrombophlebitis migrans

Thrombophlebitis neonatal

Thrombosed varicose vein

Thrombosis corpora cavernosa

Transverse sinus thrombosis

Vascular graft

Vena cava embolism

Vena cava filter insertion

Vena cava filter removal

Vena cava thrombosis



Paget-Schroetter syndrome

Pelvic venous thrombosis

Venoocclusive disease

Penile vein thrombosis

Venoocclusive liver disease

Peripheral vein occlusion Venous angioplasty

Peripheral vein thrombosis

Peripheral vein thrombus extension Venous occlusion
Phlebectomy Venous operation
Portal vein cavernous transformation Venous recanalisation

Portal vein embolism Venous repair

Portal vein occlusion Venous stent insertion
Portal vein thrombosis Venous thrombosis

Portosplenomesenteric venous thrombosis Venous thrombosis in pregnancy

Post procedural pulmonary embolism

Post thrombotic syndrome

Postoperative thrombosis

Venous thrombosis limb

Venous thrombosis neonatal

Visceral venous thrombosis

Postpartum venous thrombosis

# 8.4.2.8. Cardiac Rhythm Disturbances

The Cardiac rhythm disturbances search definition is based on the MedDRA version 27.0 Narrow and Broad Terms from the Arrhythmia related investigations, signs and symptoms SMQ. The PTs are shown below, with Narrow search terms indicated:

Chronotropic incompetence<sup>1</sup> Electrocardiogram ambulatory abnormal

Early repolarisation syndrome<sup>1</sup>

Electrocardiogram repolarisation Electrocardiogram change

abnormality<sup>1</sup>

Electrocardiogram RR interval abnormal<sup>1</sup>

Electrocardiogram RR interval prolonged<sup>1</sup> Heart rate abnormal

Electrocardiogram RR interval shortened<sup>1</sup>

Electrocardiogram U wave inversion<sup>1</sup> Heart rate decreased
Electrocardiogram U wave present<sup>1</sup> Heart rate increased
Electrocardiogram U-wave abnormality<sup>1</sup> Loss of consciousness

Sudden cardiac death<sup>1</sup> Palpitations

Bezold-Jarisch reflex Rebound tachycardia

Bradycardia Respiratory sinus arrhythmia magnitude

abnormal

Cardiac arrest Respiratory sinus arrhythmia magnitude

decreased

Cardiac death Respiratory sinus arrhythmia magnitude



increased

Cardiac telemetry abnormal
Cardio-respiratory arrest
Central bradycardia
Sudden death
Syncope
Tachycardia

Cerebrocardiac syndrome

Electrocardiogram abnormal Tachycardia paroxysmal

# 8.4.2.9. Upper Respiratory Tract Infections

The Upper respiratory tract infections search definition based on the following selected MedDRA version 27.0 PTs:

Acute sinusitis Sinusitis

Upper respiratory tract infection Viral upper respiratory tract infection

#### 8.4.2.10. Diarrhea

The Diarrhea search definition is based on the MedDRA version 27.0 PT of Diarrhoea.

<sup>&</sup>lt;sup>1</sup>Narrow term



# **Plan Version History**

| Version | Effective Date | Changes | Author / Modified by |
|---------|----------------|-------------------|----------------------|
| 1.0 | 17-Feb-2023 | NA | Steven Chang |
| 2.0 | 03-Jun-2024 | See summary below | Eve Zeng |
| 3.0 | 28-Oct-2024 | See summary below | Steven Chang |

# **Change History Summary**

| Version | Modifications |
|---|---|
| 1.0 | Initial Version |
| 2.0 | PFS-6 was redefined as a survival probability for consistency with the Kaplan-Meier methodology which was intended to be used to estimate this endpoint. |
| 2.0 | Definitions and analysis methods were added for PFS and OS. |
| 2.0 | Progression-free survival on continued nirogacestat treatment and PFS2 were added due to protocol amendment. |
| 2.0 | Miscellaneous formatting and typographical changes. |
| 2.0 | Statement was added for why the planned interim assessment using Bayesian approach as mentioned in the protocol was not performed. |
| 2.0 | Analysis of safety topics of special interest identified using standardized MedDRA queries (SMQ) or customized MedDRA queries was added. |
| 3.0 | Section 5.6.2 - Added a summary table for serious TEAEs by maximum severity (Grade) |
| 3.0 | Section 5.6.6 - Rows for the worst post-baseline change from baseline added to the ECG summary table. |
| 3.0 | Section 5.6.7 - Rows for the worst post-baseline change from baseline added to the vital signs summary table. |
| 3.0 | Section 8.4.1.4 Electrolyte disorder PTs were revised. Added new electrolyte disorder analyses (summary table and shift table). |

#### **Certificate Of Completion**

Envelope Id: 40641299A5654F08AF98E3810FA56FF4

Subject: Complete with Docusign: NIR-OGT-201 SAP V3.0 28Oct2024.pdf

Source Envelope:

Document Pages: 100 Certificate Pages: 5

AutoNav: Enabled

**Envelopeld Stamping: Disabled** 

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Signatures: 4

Initials: 0

Envelope Originator: Carmelita Alvero 100 Washington Blvd

5th Floor

Stamford, CT 06902

Status: Completed

Carmelita.Alvero@springworkstx.com

IP Address: 67.172.33.189

Sent: 29-Oct-2024 | 10:37

Viewed: 29-Oct-2024 | 10:37

Signed: 29-Oct-2024 | 10:38

Sent: 29-Oct-2024 | 10:37

Viewed: 31-Oct-2024 | 09:58

Signed: 31-Oct-2024 | 09:59

**Record Tracking** 

Status: Original

29-Oct-2024 | 10:33

Holder: Carmelita Alvero

Carmelita.Alvero@springworkstx.com

**Timestamp** 

Location: DocuSign

**Signer Events** Carmelita Alvero

carmelita.alvero@springworkstx.com Security Level: Email, Account Authentication

(Required)

Signature

Carmelita Alvero

Signature Adoption: Pre-selected Style

Signature ID:

FC9A7027-5907-4B62-B0EB-8FAC79DE2641

Using IP Address: 67.172.33.189

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab): I am the author of this document

**Electronic Record and Signature Disclosure:** 

Accepted: 01-Aug-2024 | 14:42

ID: 25522793-fb19-42f2-8369-ab6b459feb43

Jocelyn Lewis

Jocelyn.Lewis@springworkstx.com

**Medical Director** 

SpringWorks Therapeutics

Security Level: Email, Account Authentication

(Required)

Joulyn Lewis

Signature Adoption: Pre-selected Style

Signature ID:

D920FBC6-135E-4F3A-9DE7-358EDE3C6954

Using IP Address: 73.29.111.66

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Not Offered via DocuSign

| Signer Events | Signature | Timestamp |
|---|---|---|
| Steven Chang<br>steven.chang@springworkstx.com<br>Security Level: Email, Account Authentication<br>(Required) | Steven Chang Signature Adoption: Pre-selected Style Signature ID: | Sent: 29-Oct-2024 10:37<br>Viewed: 29-Oct-2024 10:41<br>Signed: 29-Oct-2024 10:42 |
| | 32411558-E40F-490F-83BD-132F2BF65799 Using IP Address: 172.190.184.114 With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I am the author of this document | |
| Electronic Record and Signature Disclosure:<br>Accepted: 29-Oct-2024 10:41<br>ID: 91c140c9-c50c-4722-82f2-903c52d27f7f | | |
| Steven Hege Steven.Hege@springworkstx.com Interim Head of Biometrics | Stuen Hige | Sent: 29-Oct-2024 10:37<br>Viewed: 31-Oct-2024 11:42<br>Signed: 31-Oct-2024 11:42 |
| Security Level: Email, Account Authentication (Required) | Signature Adoption: Pre-selected Style Signature ID: C5756967-5377-4E0D-AFD1-AB6D72356E5C Using IP Address: 50.47.98.13 With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document | |
| Electronic Record and Signature Disclosure:<br>Not Offered via DocuSign | | |
| In Person Signer Events | Signature | Timestamp |
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |

**Timestamps** 

29-Oct-2024 | 10:37

31-Oct-2024 | 11:42

31-Oct-2024 | 11:42

31-Oct-2024 | 11:42

**Timestamps** 

Status

Status

Hashed/Encrypted

Security Checked

Security Checked

Security Checked

**Envelope Summary Events** 

**Electronic Record and Signature Disclosure** 

Envelope Sent

Completed

Certified Delivered

Signing Complete

Payment Events

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, SpringWorks Therapeutics - Part 11 (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

## Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### **How to contact SpringWorks Therapeutics - Part 11:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: dom.reigle@springworkstx.com

#### To advise SpringWorks Therapeutics - Part 11 of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at dom.reigle@springworkstx.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

### To request paper copies from SpringWorks Therapeutics - Part 11

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to dom.reigle@springworkstx.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with SpringWorks Therapeutics - Part 11

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to dom.reigle@springworkstx.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

#### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify SpringWorks Therapeutics Part 11 as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by SpringWorks Therapeutics Part 11 during the course of your relationship with SpringWorks Therapeutics Part 11.